IND: Number: 103245 Regeneron Pharmaceuticals, Inc.

EudraCT: 2017-004921-33

**Medical/Study Director:** 

### **Clinical Study Protocol**

A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to **Evaluate the Effects of Fasinumab on Peripheral Nerve Function in Patients** with Pain due to Osteoarthritis of the Hip or Knee

**Fasinumab** Compound:

**Clinical Phase:** 2

**Protocol Number:** R475-OA-1758

**Protocol Version:** R475-OA-1758 Amendment 2

**Amendment 2 Date of Issue:** See appended electronic signature page

**Amendment 1 Date of Issue:** 16 Jul 2018

**Original Date of Issue** 20 Feb 2018

Regeneron Pharmaceuticals, Inc. 777 Old Saw Mill River Road

Tarrytown, NY 10591



### AMENDMENT HISTORY

### **Amendment 2**

The purpose of this amendment is to revise the criterion for detecting a change in nerve conduction velocity that would be considered not to be within established parameters, in order to reduce false-positive findings. Additional minor changes have been made to improve clarity. The following table outlines the changes made to the protocol and the affected sections:

| Change and Rationale | Sections Changed |
|---|---|
| Main Change: | |
| The criterion for detection of a change in nerve conduction velocity has been revised from a deficit of 5 m/second to a deficit of >12% relative to the baseline value. This update was made to allow the measurement of change from baseline to be relative to the patient's size (eg, height and length of limb) and, thus, decrease the potential of obtaining false-positive findings due to varying patient size. Procedures for monitoring peripheral sensory adverse events of special interest have been updated accordingly. | Section 9.6.1.3 Peripheral Sensory Adverse Events |
| Other Changes: | |
| Time frames have been added to the safety endpoints for clarity. | Clinical Study Protocol Synopsis, Endpoints Section 4.3 Additional Safety Endpoints |
| Text has been updated to align with current best practices (ie, updated protocol template text) | Clinical Study Protocol Synopsis, Endpoints Section 4.5 Anti-Drug Antibody Variables Section 10.3.4 Anti-Drug Antibody Analysis Set Section 10.4.6 Analysis of Anti-Drug Antibody Data Section 14.5 Clinical Study Data Transparency (section added) |
| An additional reason for permanent discontinuation of study drug has been added, as follows: 'Per protocol repeated nerve conduction test that confirms results are not within the established parameters for peroneal, sural, or ulnar nerves, as per central reader assessment and the neurologist's evaluation that confirms the diagnosis of peripheral neuropathy.' | Section 7.3.2.1 Reasons for Permanent Discontinuation of Study Drug |

| Minor edits were also made to this section. | |
|---|---|
| A statement has been added to clarify that patient- | Table 1 Schedule of Events |
| reported outcome measures should be completed before all other assessments. | Section 8.1.1 Footnotes for the Schedule of Events Table 1, Footnote #22 |
| | Section 8.2.2.1 Western Ontario and McMaster Universities Osteoarthritis Index |
| | Section 8.2.3.3 Survey of Autonomic Symptoms |
| | Section 8.2.4.4 Joint Pain Questionnaire |
| Methotrexate has been added to the list of prohibited immunosuppressants. | Section 7.7.1 Prohibited Medications |
| The scale used to assess the WOMAC index has been revised to the numerical rating scale (previously incorrectly cited as the Likert scale). | Section 8.2.2.1 Western Ontario and McMaster Universities Osteoarthritis Index |
| RAVE Medidata Imaging System has been added to the list of electronic systems used in the study. This is an electronic platform used to upload nerve conduction test wave forms for central reader review. | Section 11.2 Electronic Systems |
| Other edits have been made throughout the document to | Clinical Study Protocol Synopsis, Study Design |
| improve clarity or correct minor errors. | List of Abbreviations and Definition of Terms |
| | Section 5.1.1 Screening and Pre-Randomization |
| | Section 5.1.2 Rescreening |
| | Section 6.2.2 Exclusion Criteria, #7 |
| | Section 7.1 Investigational and Reference Treatments |
| | Section 7.3.2.2 Reasons for Temporary Discontinuation of Study Drug |
| | Table 1 Schedule of Events |
| | Section 8.1.1 Footnotes for the Schedule of Events Table 1, Footnote #8, Footnote #19 |
| | Section 8.2.3.1 Nerve Conduction |
| | Section 8.2.4.8 Laboratory Testing |
| | Section 10.4.5 Analysis of Drug Concentration Data |

### Amendment 1

The purpose of this amendment is to change the fasinumab 3 mg Q4W dose regimen to a 1 mg Q4W dose regimen because the 3 mg Q4W dose regimen is no longer being evaluated in the osteoarthritis (OA) pain program. The 1 mg Q4W dose regimen is now the highest dose being evaluated in this patient population. Additional changes have been made to improve study outcome measures and for clarity. The following table outlines the changes made to the protocol and the affected sections:

| Change and Rationale | Sections Changed |
|---|---|
| The 3 mg Q4W dose regimen has been removed and replaced with a 1 mg Q4W dose regimen. | Clinical Study Protocol Synopsis, Study Design,<br>Treatments, Statistical Plan |
| | Section 1 Introduction |
| | Section 3.1.2 Rationale for Dose Selection |
| | Section 5.1.3 Randomization |
| | Section 5.1.4 Treatment Period |
| | Section 7.1 Investigational and Reference Treatments |
| | Section 7.5 Method of Treatment Assignment |
| | Section 10.2 Justification of Sample Size |
| The phone visit at week 1 has been changed to a site visit in order to obtain a more complete pharmacokinetic profile. | Table 1 Schedule of Events |
| The exclusion criterion regarding carpal tunnel syndrome has been updated to include additional conditions that could interfere with the assessment of the primary endpoint. Specifically, "Signs or symptoms of carpal tunnel syndrome within 6 months of the screening visit" has been updated to "History or presence of signs or symptoms of compression neuropathy, including carpal tunnel syndrome or sciatica." | Section 6.2.2 Exclusion Criteria, #4 |
| Text has been added to clarify that the results of the nerve conduction assessment must be obtained before randomization can occur. | Clinical Study Protocol Synopsis, Study Design Section 5.1.1 Screening and Pre-Randomization Table 1 Schedule of Events Section 8.1.1 Footnotes for the Schedule of Events, Table 1 Footnote #8 |
| Drugs included in the urine drug test have been listed in<br>the Laboratory Testing section | Section 8.2.4.8 Laboratory Testing |

Additional text has been added, edited or deleted in order to improve clarity of the protocol, to make minor corrections, to be consistent across fasinumab program, or to align with current Regeneron best practices.

Clinical Study Protocol Synopsis, Safety Endpoints

List of Abbreviations and Definitions of Terms

Section 4.3 Additional Safety Endpoints

Section 5.1.1 Screening and Pre-Randomization

Section 5.1.2 Rescreening

Section 6.2.2 Exclusion Criteria, #7

Section 7.4.2 Local Injection Site Reactions

Section 7.7.1 Prohibited Medications

Section 7.7.2 Permitted Medications and Procedures

Table 1, Schedule of Events

Section 8.1.1 Footnotes for the Schedule of Events

Table 1, Footnote #4

Section 8.2.1.8 Diary Training

Section 8.2.1.9 Patient Education Brochures

Section 8.2.4.7 Procedures to be Performed Only in the

Event of a Joint Replacement Surgery

Section 9.4.3 Other Events that Require Accelerated

Reporting to Sponsor

Section 9.6.1.1 Adjudicated Arthropathy

Section 9.6.1.3 Peripheral Sensory Adverse Events

Section 10.3.3 Pharmacokinetic Analysis Set

Section 10.4.3 Efficacy Analysis

Section 10.4.5 Analysis of Drug Concentration Data

Section 11.2 Electronic Systems

Section 12.1 Monitoring of Study Sites

### **TABLE OF CONTENTS**

| CLINIC | AL STUDY PROTOCOL SYNOPSIS | 12 |
|--------|---------------------------------------------------|----|
| LIST O | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 18 |
| 1. | INTRODUCTION | 20 |
| 2. | STUDY OBJECTIVES | 23 |
| 2.1. | Primary Objective | 23 |
| 2.2. | Secondary Objectives | 23 |
| 3. | RATIONALE | 24 |
| 3.1. | Rationale | 24 |
| 3.1.1. | Rationale for Study Design | 24 |
| 3.1.2. | Rationale for Dose Selection | 24 |
| 4. | STUDY VARIABLES | 25 |
| 4.1. | Demographic and Baseline Characteristics | 25 |
| 4.2. | Primary and Secondary Endpoints | 25 |
| 4.2.1. | Primary Endpoints | 25 |
| 4.2.2. | Secondary Endpoints | 25 |
| 4.3. | Additional Safety Endpoints | 25 |
| 4.4. | Pharmacokinetic Variables | 26 |
| 4.5. | Anti-Drug Antibody Variables | 26 |
| 5. | STUDY DESIGN | 26 |
| 5.1. | Study Description and Duration | 26 |
| 5.1.1. | Screening and Pre-Randomization | 26 |
| 5.1.2. | Rescreening | 27 |
| 5.1.3. | Randomization | 28 |
| 5.1.4. | Treatment Period | 28 |
| 5.1.5. | Follow-up Period | 28 |
| 5.1.6. | End of Study Phone Contact and Additional Imaging | 28 |
| 5.1.7. | Study Stopping Rules | 28 |
| 5.1.8. | End of Study Definition. | 29 |
| 5.2. | Planned Interim Analysis. | 29 |
| 5.3. | Study Committees | 29 |
| 5.3.1. | Independent Data Monitoring Committee | 29 |

| 5.3.2. | Arthropathy Adjudication Committee | 29 |
|----------|-------------------------------------------------------------|----|
| 6. | SELECTION, WITHDRAWAL, AND REPLACEMENT OF PATIENTS | 29 |
| 6.1. | Number of Patients Planned | 29 |
| 6.2. | Study Population | 30 |
| 6.2.1. | Inclusion Criteria | 30 |
| 6.2.2. | Exclusion Criteria | 31 |
| 6.3. | Premature Withdrawal from the Study | 34 |
| 6.4. | Replacement of Patients | 35 |
| 7. | STUDY TREATMENTS | 35 |
| 7.1. | Investigational and Reference Treatments | 35 |
| 7.2. | Rescue Treatment | 35 |
| 7.3. | Dose Modification and Study Treatment Discontinuation Rules | 36 |
| 7.3.1. | Dose Modification | 36 |
| 7.3.2. | Study Drug Discontinuation | 36 |
| 7.3.2.1. | Reasons for Permanent Discontinuation of Study Drug | 36 |
| 7.3.2.2. | Reasons for Temporary Discontinuation of Study Drug | 38 |
| 7.4. | Management of Acute Reactions | 38 |
| 7.4.1. | Systemic Injection Reactions. | 38 |
| 7.4.2. | Local Injection Site Reactions | 38 |
| 7.5. | Method of Treatment Assignment | 38 |
| 7.5.1. | Blinding | 38 |
| 7.5.2. | Emergency Unblinding | 39 |
| 7.5.3. | Unblinding for Regulatory Reporting Purposes | 39 |
| 7.6. | Treatment Logistics and Accountability | 39 |
| 7.6.1. | Packaging, Labeling, and Storage | 39 |
| 7.6.2. | Supply and Disposition of Treatments | 39 |
| 7.6.3. | Treatment Accountability | 40 |
| 7.6.4. | Treatment Compliance. | 40 |
| 7.7. | Concomitant Medications and Procedures | 40 |
| 7.7.1. | Prohibited Medications | 40 |
| 7.7.2. | Permitted Medications and Procedures | 41 |
| 8. | STUDY SCHEDULE OF EVENTS AND PROCEDURES | 41 |
| 8.1. | Schedule of Events | 41 |

| 8.1.1. | Footnotes for the Schedule of Events Table 1 | 45 |
|---|---|---|
| 8.1.2. | Footnotes for Table 2 - Follow-up Period for Patients Undergoing Joint Replacement Surgery | 47 |
| 8.1.3. | Early Termination Visit | 48 |
| 8.1.4. | Unscheduled Visits | 48 |
| 8.2. | Study Procedures | 48 |
| 8.2.1. | Procedures Performed Only at the Screening/Baseline Visit | 48 |
| 8.2.1.1. | Main Study Informed Consent | 48 |
| 8.2.1.2. | Genomics Sub-study Informed Consent | 48 |
| 8.2.1.3. | Medical History | 48 |
| 8.2.1.4. | Medication History | 48 |
| 8.2.1.5. | Demographics | 49 |
| 8.2.1.6. | Determination of Osteoarthritis | 49 |
| 8.2.1.7. | Assessment of Childbearing Potential | 49 |
| 8.2.1.8. | Diary Training | 50 |
| 8.2.1.9. | Patient Education Brochures | 50 |
| 8.2.2. | Patient-Completed Assessments and Efficacy Procedures | 50 |
| 8.2.2.1. | Western Ontario and McMaster Universities Osteoarthritis Index | 50 |
| 8.2.3. | Neurological Assessments | 50 |
| 8.2.3.1. | Nerve Conduction | 50 |
| 8.2.3.2. | Neurological Examination (Full) | 51 |
| 8.2.3.3. | Survey of Autonomic Symptoms | 51 |
| 8.2.3.4. | Orthostatic Blood Pressure Assessment and Heart Rate | 51 |
| 8.2.4. | Safety Procedures | 52 |
| 8.2.4.1. | Vital Signs | 52 |
| 8.2.4.2. | Electrocardiogram | 52 |
| 8.2.4.3. | Physical Examination and Body Weight | 52 |
| 8.2.4.4. | Joint Pain Questionnaire | 52 |
| 8.2.4.5. | Imaging | 52 |
| 8.2.4.6. | End of Study Phone Contact and Additional Imaging | 53 |
| 8.2.4.7. | Procedures to be Performed Only in the Event of a Joint Replacement Surgery | 53 |
| 8.2.4.8. | Laboratory Testing | |

| 8.2.4.9. | Injection Site Evaluations | 56 |
|---|---|---|
| 8.2.5. | Pharmacokinetic and Anti-Drug Antibody Procedures | 56 |
| 8.2.5.1. | Drug Concentration Measurements and Samples | 56 |
| 8.2.5.2. | Anti-Drug Antibody Measurements and Samples | 56 |
| 8.2.6. | Research Samples | 56 |
| 8.2.6.1. | Biomarkers | 56 |
| 8.2.6.2. | Future Biomedical Research | 57 |
| 8.2.6.3. | Genomics Sub-study - Optional | 57 |
| 9. | SAFETY DEFINITIONS, REPORTING, AND MONITORING | 58 |
| 9.1. | Obligations of Investigator | 58 |
| 9.2. | Obligations of Sponsor | 58 |
| 9.3. | Definitions | 58 |
| 9.3.1. | Adverse Event | 58 |
| 9.3.2. | Serious Adverse Event | 58 |
| 9.3.3. | Adverse Events of Special Interest | 59 |
| 9.4. | Recording and Reporting Adverse Events | 59 |
| 9.4.1. | Adverse Events | 59 |
| 9.4.2. | Serious Adverse Events | 59 |
| 9.4.3. | Other Events that Require Accelerated Reporting to Sponsor | 60 |
| 9.4.4. | Reporting Adverse Events Leading to Withdrawal from the Study | 61 |
| 9.4.5. | Abnormal Laboratory, Vital Signs, or Electrocardiogram Results | 61 |
| 9.4.6. | Follow-up | 61 |
| 9.5. | Evaluation of Severity and Causality | 61 |
| 9.5.1. | Evaluation of Severity | 61 |
| 9.5.2. | Evaluation of Causality | 62 |
| 9.6. | Safety Monitoring | 64 |
| 9.6.1. | Monitoring Adverse Events of Special Interest | 64 |
| 9.6.1.1. | Adjudicated Arthropathy | 64 |
| 9.6.1.2. | Sympathetic Nervous System Dysfunction | 65 |
| 9.6.1.3. | Peripheral Sensory Adverse Events | 66 |
| 9.6.1.4. | Joint Replacement Surgery | 66 |
| 9.7. | Investigator Alert Notification | 67 |
| 10. | STATISTICAL PLAN | 67 |

| 10.1. | Statistical Hypothesis | 67 |
|---|---|---|
| 10.2. | Justification of Sample Size | 67 |
| 10.3. | Analysis Sets | 68 |
| 10.3.1. | Efficacy Analysis Set | 68 |
| 10.3.2. | Safety Analysis Set | 68 |
| 10.3.3. | Pharmacokinetic Analysis Set | 68 |
| 10.3.4. | Anti-Drug Antibody Analysis Set | 68 |
| 10.4. | Statistical Methods | 68 |
| 10.4.1. | Patient Disposition | 68 |
| 10.4.2. | Demography and Baseline Characteristics | 68 |
| 10.4.3. | Efficacy Analysis | 69 |
| 10.4.4. | Safety Analysis | 69 |
| 10.4.4.1. | Primary Safety Analysis | 69 |
| 10.4.4.2. | Adverse Events | 70 |
| 10.4.4.3. | Other Safety | 70 |
| 10.4.4.4. | Treatment Exposure | 71 |
| 10.4.4.5. | Treatment Compliance. | 71 |
| 10.4.5. | Analysis of Drug Concentration Data. | 71 |
| 10.4.6. | Analysis of Anti-Drug Antibody Data | 71 |
| 10.5. | Interim Analysis | 72 |
| 10.6. | Additional Statistical Data Handling Conventions | 72 |
| 10.7. | Statistical Considerations Surrounding the Premature Termination of a Study | 72 |
| 11. | DATA MANAGEMENT AND ELECTRONIC SYSTEMS | 73 |
| 11.1. | Data Management | 73 |
| 11.2. | Electronic Systems. | 73 |
| 12. | STUDY MONITORING | 73 |
| 12.1. | Monitoring of Study Sites | 73 |
| 12.2. | Source Document Requirements | 73 |
| 12.3. | Case Report Form Requirements | 74 |
| 13. | AUDITS AND INSPECTIONS | 74 |
| 14. | ETHICAL AND REGULATORY CONSIDERATIONS | 75 |
| 14.1. | Good Clinical Practice Statement | 75 |
| 14.2. | Informed Consent | 75 |

| 14.3. | Patient Confidentiality and Data Protection | 75 |
|---|---|---|
| 14.4. | Institutional Review Board/Ethics Committee | 76 |
| 14.5. | Clinical Study Data Transparency | 76 |
| 15. | PROTOCOL AMENDMENTS | 76 |
| 16. | PREMATURE TERMINATION OF THE STUDY OR CLOSE-OUT OF A SITE | 76 |
| 16.1. | Premature Termination of the Study | 76 |
| 16.2. | Close-out of a Site | 76 |
| 17. | STUDY DOCUMENTATION | 77 |
| 17.1. | Certification of Accuracy of Data. | 77 |
| 17.2. | Retention of Records | 77 |
| 18. | DATA QUALITY ASSURANCE | 77 |
| 19. | CONFIDENTIALITY | 78 |
| 20. | FINANCING AND INSURANCE | 78 |
| 21. | PUBLICATION POLICY | 78 |
| 22. | REFERENCES | 79 |
| 23. | INVESTIGATOR'S AGREEMENT | 82 |
| SIGNATU | JRE OF SPONSOR'S RESPONSIBLE OFFICERS | 83 |
| | LIST OF TABLES | |
| Table 1: | Schedule of Events | 42 |
| Table 2: | Follow-up Period for Patients Undergoing Joint Replacement Surgery on Study | 47 |
| | LIST OF FIGURES | |
| Figure 1: | Study Flow Diagram | 26 |

### CLINICAL STUDY PROTOCOL SYNOPSIS

| CLINIC | AL STUDY PROTOCOL SYNOPSIS |
|---|---|
| Title | A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to<br>Evaluate the Effects of Fasinumab on Peripheral Nerve Function in Patients<br>with Pain Due to Osteoarthritis of the Hip or Knee |
| Site Locations | To be determined. |
| Principal Investigator | |
| Objectives | Primary Objective |
| | The primary objective of the study is to evaluate the effect of fasinumab compared to placebo on peripheral nerves in patients with pain due to osteoarthritis (OA) of the hip or knee. |
| | Secondary Objectives |
| | The secondary objectives of the study are: |
| | • To evaluate the efficacy of fasinumab compared to placebo in patients with pain due to OA of the hip or knee |
| | To evaluate the safety and tolerability of fasinumab compared to<br>placebo in patients with pain due to OA of the hip or knee |
| | • To characterize the concentrations of fasinumab in serum in patients with pain due to OA of the hip or knee |
| | • To evaluate the immunogenicity of fasinumab in patients with pain due to OA of the hip or knee |
| Study Design | This is a phase 2, randomized, double-blind, placebo-controlled, multicenter study designed to evaluate the neurological safety of fasinumab compared to placebo in patients with pain due to OA of the hip or knee. In addition, the safety, efficacy, pharmacokinetics (PK), and immunogenicity of fasinumab compared to placebo will be assessed. |
| | The study duration will be approximately 64 weeks starting at randomization (day 1). The study consists of a screening period of up to 30 days, a 7 to 10 day pre-randomization period (7 days with a +3 day window), a 16-week treatment period (with the last every 4 week [Q4W] dose of study drug administered at week 12), a 20-week follow-up period, and a final phone contact approximately 52 weeks after the last dose of study drug is administered. |
| | Screening and Pre-Randomization |
| | Prior to randomization, patients will undergo screening procedures, including X-ray of the shoulders, hips, and knees. Magnetic resonance imaging (MRI) of the index and contralateral joints must be performed at |

Regeneron Pharmaceuticals, Inc.


screening and the results assessed by the central imaging vendor. In addition, an MRI will be performed on any knee or hip joint with a Kellgren-

Lawrence (K-L) score of ≥3. Randomization visits cannot occur until there is confirmation from the central imaging vendor that there are no exclusionary findings on the X-rays and any required MRIs.

Prior to randomization, patients will also undergo nerve conduction assessments. Patients must complete all other inclusion/exclusion assessments before undergoing the nerve conduction assessments. Randomization cannot occur until there is confirmation from the central reader assessment that the results are within the established parameters.

During the screening period, patients may continue to take their current treatment regimen for OA pain.

Patients eligible for the study will complete a pre-randomization period. The pre-randomization visit will be 7 to 10 days before the randomization visit. During this period, patients will discontinue and/or undergo a washout of their current pain medications for OA. All pain medication, except for the study-provided rescue medication (acetaminophen/paracetamol), will be discontinued.

#### Randomization

On day 1 (baseline), approximately 180 patients will be randomized in a 1:1 ratio to fasinumab 1 mg subcutaneous (SC) Q4W or fasinumab-matching placebo SC Q4W. Randomization will be stratified according to the affected index joint (hip or knee) and the K-L score (2 to 3, or 4) at the screening visit.

#### **Treatment**

During the treatment period (day 1 through week 16), patients will be permitted to use only study-provided acetaminophen/paracetamol as rescue medication. Patients will record their use of acetaminophen/paracetamol in a diary.

Neurological, efficacy and safety assessments will be performed during the treatment period.

#### Follow-up

Follow-up of patients will continue for an additional 20 weeks after the last treatment period visit. Neurological, efficacy, and safety assessments will be performed during this period.

If a patient must undergo joint replacement (JR) surgery during the follow-up period, he or she will be asked to complete pre-operative imaging and to undergo post-surgery follow-up.

#### **End of study Phone Contact**

A phone contact questionnaire will be conducted at approximately 52 weeks after administration of the last dose of study drug to document patient status with regard to JR surgery (if patient underwent, is scheduled for, or is on a

| | wait list for JR surgery). Patients who had an adjudicated arthropathy (AA) will have an MRI performed of the affected joint(s). |
|---|---|
| Study Duration | The duration of the study is up to 64 weeks, excluding the screening and pre-randomization periods. Patients who discontinue study drug will be requested to return for all scheduled study visits and to complete all planned assessments, including phone contacts. |
| End of Study Definition | The end of study is defined as the last phone contact of the last patient in this study. |
| Population | |
| Sample Size: | Enrollment of approximately 180 patients is planned for this study (approximately 90 patients per treatment group) |
| Target Population: | Men and women who are at least 18 years of age at the time of study entry with a clinical diagnosis at the screening visit of OA of the knee or hip, based on the American College of Rheumatology criteria, and with radiologic evidence of OA (K-L score ≥2) at the index joint. |
| Treatments | |
| Study Drug Dose/Route/Schedule: | Fasinumab 1 mg SC Q4W |
| Study Drug Placebo Route/Schedule: | Fasinumab-matching placebo<br>SC Q4W |
| Rescue Treatment: | Starting at pre-randomization to the end of the 16-week treatment period, acetaminophen/paracetamol is the only study-provided rescue medication. In the event of inadequate pain relief for OA or in the event of other pain (eg, headache) or fever, 1 to 2 tablets/capsules of acetaminophen/paracetamol may be taken no less than 4 hours apart as needed according to the local standard of care. |
| Endpoints | |
| Primary: | The primary endpoints of the study are: |
| | <ul> <li>Change from baseline to week 16 in peroneal motor nerve<br/>conduction velocity</li> </ul> |
| | <ul> <li>Change from baseline to week 16 in peroneal motor nerve action<br/>potential amplitude</li> </ul> |
| | Change from baseline to week 16 in sural sensory nerve conduction velocity |
| | <ul> <li>Change from baseline to week 16 in sural sensory nerve action<br/>potential amplitude</li> </ul> |

- Change from baseline to week 16 in ulnar sensory nerve conduction velocity
- Change from baseline to week 16 in ulnar sensory nerve action potential amplitude

#### **Secondary:**

The secondary endpoints of the study are:

- Change from baseline to week 16 in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score
- Change from baseline to week 16 in WOMAC physical function subscale score

#### Safety:

Additional safety endpoints in this study include:

- Incidence of AA (as confirmed by an independent adjudication committee) through week 36
- Incidence of destructive arthropathy (DA) (as confirmed by an independent adjudication committee) through week 36
- Incidence of treatment-emergent adverse event (TEAEs) through week 16
- Incidence of sympathetic nervous system (SNS) dysfunction (as diagnosed after consultation with an appropriate specialist, such as a neurologist and/or cardiologist) through week 36
- Incidence of peripheral sensory adverse events (AEs) that require a neurology or other specialty consultation through week 36
- Incidence of all-cause JR surgeries through week 36
- Incidence of JRs at telephone survey approximately 52 weeks after last dose of study drug

# Pharmacokinetic variable:

The PK variable is the concentration of functional fasinumab in serum samples collected at specified time points.

## Anti-drug antibody variables:

Anti-drug antibody (ADA) variables include status (positive or negative), titer, and time point/visit.

#### **Procedures and Assessments**

At the screening visit, patients will provide informed consent, medical history, and medication history. Determination of the K-L score of the knee or hip will be performed to establish a diagnosis of OA based on the American College of Rheumatology criteria using a K-L score cutoff of ≥2. Patients will be assessed for childbearing potential.

### Regeneron Pharmaceuticals, Inc.

Peripheral nerve function will be assessed by measuring nerve conduction velocities and evoked amplitudes of the peroneal motor, sural sensory and ulnar sensory nerves.

Additional safety assessments will be performed at each study visit and upon occurrence of any joint AEs. Potential events of AA will be monitored via clinical signs and symptoms of worsening joint pain during the study and adjudication of pre-operative imaging for patients who undergo JR during the conduct of the study. Potential events of SNS dysfunction will be monitored throughout the study through physical examination, AE reporting, assessment of orthostatic hypotension, and the Survey of Autonomic Symptoms.

Efficacy will be assessed using WOMAC pain and physical function subscale scores.

Approximately 52 weeks after administration of the last study dose, a phone contact questionnaire will be conducted to document patient status with regard to JR surgery (if patient underwent, is scheduled for, or is on a wait list for JR surgery). Patients who had an AA will have an MRI performed of the affected joint(s).

#### Statistical Plan

#### **Statistical Hypothesis**

No formal hypothesis testing will be performed on nerve conduction measures. The treatment difference between fasinumab and placebo in the change from baseline to week 16 in nerve conduction measures will be estimated and presented descriptively along with 95% confidence intervals.

#### **Justification of Sample Size**

Approximately 180 patients will be randomized in a 1:1 ratio to fasinumab 1 mg Q4W or placebo. With this sample size, the precision of the estimated treatment difference between fasinumab and placebo at week 16 in nerve conduction velocity is no more than 1.21 m/s with a 95% confidence level, assuming a standard deviation (SD) of 3.6 m/s. This sample size provides similar precision for the estimated treatment difference in nerve conduction amplitude assuming a SD of 3.6  $\mu$ V. Assuming a 2-sided alpha level of 0.05 and a 15% dropout rate up to week 16, an enrollment of 90 patients per group will provide at least 80% power to detect an effect size of 0.46 in the WOMAC pain and physical function subscale scores (ie, absolute treatment difference of 1.1 between fasinumab and placebo with an SD of 2.4). The assumed treatment difference and SD are based on results from study R475-PN-1227.

#### **Statistical Methods**

For continuous variables, descriptive statistics will include the following information: the number of patients reflected in the calculation (n), mean, median, standard deviation, minimum, Q1, Q3, and maximum.

For categorical or ordinal data, frequencies and percentages will be displayed for each category.

Safety data including nerve conduction measures, TEAEs and treatmentemergent adverse events of special interest (AESIs), vital signs, physical exams, laboratory tests, electrocardiograms (ECGs), and ADA formation will be listed and summarized by treatment group. The nerve conduction variables will be analyzed using a mixed-effect model repeated measure (MMRM) approach based on the safety analysis set (SAF). The leastsquares mean estimates for the mean change from baseline to week 16, as well as the differences of the estimates between fasinumab and placebo, with their corresponding standard errors and associated 95% confidence intervals, will be provided descriptively.

The efficacy variables will be analyzed using multiple imputation approach with MMRM based on the full analysis set (FAS) with adjustment for missing data due to lack of efficacy or AEs assuming the scores would on average return to baseline values.

For analysis of categorical variables, eg, proportions of patients with ≥30% improvement in the WOMAC pain subscale scores at week 16, the Cochran Mantel Haenszel approach stratified by the randomization strata will be used with missing data considered as non-response.

Summaries of serum concentrations of functional fasinumab will be presented by nominal time point. Plots of individual concentration over time will be presented by actual day. Plots of mean or median concentrations of functional fasinumab will be presented by nominal day. No formal statistical analysis will be performed.

### LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

5-ASA 5-aminosalicylic acid

AA Adjudicated arthropathy

ADA Anti-drug antibody

AE Adverse event

AESI Adverse event of special interest

ALT Alanine aminotransferase
AST Aspartate aminotransferase

AUC Area under the curve bpm Beats per minute

CRF Case report form (electronic or paper)

CRO Contract research organization

CTCAE Common Terminology Criteria for Adverse Events

DA Destructive arthropathy

DMC Data Monitoring Committee

EC Ethics Committee
ECG Electrocardiogram

EDC Electronic data capture

ESR Erythrocyte sedimentation rate

FAS Full analysis set

FDA Food and Drug Administration
FSH Follicle-stimulating hormone

GCP Good Clinical Practice

HbA1c Hemoglobin A1c

HIV Human immunodeficiency virus

ICF Informed consent form

ICH International Council for Harmonisation

INR International normalized ratio
IRB Institutional Review Board

IV Intravenous

IWRS Interactive web response system

JR Joint replacement
K-L Kellgren-Lawrence

MedDRA Medical Dictionary for Regulatory Activities

MMRM Mixed-effect Model for Repeated Measures

MRI Magnetic Resonance Imaging

NGF Nerve growth factor

NSAID Nonsteroidal anti-inflammatory drug

OA Osteoarthritis

PCSV Potentially clinically significant value

PK Pharmacokinetic
PT Preferred term

QRS Complex of Q, R, and S waves on an electrocardiogram

Q4W Every 4 weeks
Q8W Every 8 weeks
RBC Red blood cell

Regeneron Pharmaceuticals, Inc.

SAE Serious adverse event SAF Safety analysis set

SAP Statistical analysis plan
SAS Statistical Analysis System

SC Subcutaneous

SD Standard deviation

SNS Sympathetic Nervous System

SOC System organ class

SUSAR Suspected unexpected serious adverse reaction

TBL Total bilirubin

TEAE Treatment-emergent adverse event

TJR Total joint replacement
TrkA Tyrosine kinase type 1
ULN Upper limit of normal
WBC White blood cell

WOCBP Woman of child-bearing potential

WOMAC Western Ontario and McMaster Universities Osteoarthritis Index

#### 1. INTRODUCTION

Chronic musculoskeletal pain affects a large proportion of the global population. A significant cause of chronic musculoskeletal pain is due to osteoarthritis (OA). Osteoarthritis is a progressive, chronic disease caused by the breakdown and loss of cartilage of the joints, which leads to pain in the hips, knees, hands, feet, and spine. It is characterized by focal areas of loss of articular cartilage in synovial joints accompanied by subchondral bone changes, osteophyte formation at the joint margins, thickening of the joint capsule and mild synovitis. Symptoms and disability increase with increasing age. The prevalence of OA in patients aged 65 and older is 60% in men and 70% in women, and is continually rising (Sarzi-Puttini 2005).

Nonsteroidal anti-inflammatory drugs (NSAIDs) are the mainstay of treatment in patients with mild-to-moderate OA. The efficacy of NSAIDs is well documented, albeit modest, but their use is associated with a number of risks (Bingham 2007, Bjordal 2004, Makarowski 2002, Silverstein 2000). The risks associated with long-term therapy with NSAIDs in particular, have been well characterized and include gastrointestinal bleeding and increased risk of cardiovascular events (Lanas 2011, Trelle 2011). Nonsteroidal anti-inflammatory drugs have limited efficacy in many OA patients; those with advanced OA typically try several NSAIDs and must often escalate to other therapies such as opioids.

Treatment guidelines for OA suggest that opioids may be used in OA only if management with NSAIDs is ineffective, intolerable, or otherwise contraindicated. However, the use of opioids is limited by central nervous system effects, nausea and vomiting, constipation, and potential for abuse and dependence. In addition, opioid use may be associated with both acute and chronic side effects, including drowsiness, dizziness, gastrointestinal intolerability, motor imbalance, respiratory depression, and even death. Opioid use must be closely monitored in patients who are vulnerable or potentially vulnerable to abuse or addiction. Moreover, there is no evidence to support superiority of opioids over other available pain medications. While the efficacy of opioids in treating pain over a short duration is supported by research data, long-term efficacy has not been evaluated.

Thus, there remains an unmet medical need for alternative treatment options to opioids that have a more effective analgesic effect, particularly since there are a significant number of patients who are intolerant to or do not get adequate pain relief from the currently available treatment options. Inadequate pain relief has a profound impact on the quality of life for millions of people worldwide with an associated substantial cost to society, including healthcare cost (Salmon 2016) and loss of productivity (Dibonaventura 2011).

Neurotrophins are a family of peptide growth factors that play a role in the development, differentiation, survival, and death of neuronal and non-neuronal cells (Chao 2006). Nerve growth factor (NGF) was the first neurotrophin to be identified, and its role in the development and survival of both peripheral and central neurons during the development of the nervous system is well characterized (Crowley 1994, Smeyne 1994). In the adult, NGF is not required as a survival factor but acts as a pain mediator that sensitizes neurons (Pezet 2006). Nerve growth factor activity is mediated through 2 different membrane-bound receptors, the high-affinity tyrosine kinase type 1 (TrkA) and the low-affinity p75 neurotrophin receptors.

By acting upstream of several relevant molecular pathways, the NGF/TrkA system appears to play a major role in the control of pain. Administration of NGF has been shown to provoke pain in both

rodents (Lewin 1994) and humans (McArthur 2000), while NGF antagonists have been shown to prevent hyperalgesia and allodynia in animal models of neuropathic and chronic inflammatory pain (Ramer 1999). Humans with mutations in TrkA (hereditary sensory and autonomic neuropathy IV) or NGF (hereditary sensory and autonomic neuropathy V) have been identified with a loss of deep pain perception (Einarsdottir 2004, Indo 1996). In addition, NGF is known to be elevated in the synovial fluid of patients with rheumatoid arthritis and other types of arthritis (Aloe 1992, Halliday 1998), and to be up-regulated in injured and inflamed tissues in conditions such as cystitis, prostatitis, and chronic headache (Lowe 1997, Miller 2002, Sarchielli 2001).

Fasinumab (also known as REGN475) is a fully-human high-affinity monoclonal antibody directed against NGF. By selectively blocking NGF, fasinumab has the potential to be effective in modulating NGF-associated pain without some of the adverse side effects of other analgesic medications, such as opioids and NSAIDs. Following an evaluation of the safety and tolerability of the antibody in a single-ascending-dose first-in-human study (study R475-PN-0817), a proof-of-concept study evaluating the effect of fasinumab on pain in 217 patients with OA of the knee was completed (study R475-PN-0901, see current version of the Fasinumab Investigator's Brochure). Three intravenous (IV) doses of fasinumab were evaluated (0.03, 0.1, 0.3 mg/kg every 8 weeks [O8W]). All 3 doses, compared with placebo, were associated with statistically significant improvement in pain as evaluated by walking knee pain, the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and the Patient's Global Impression of Change questionnaire. Additionally, another study (R475-PN-1227) in patients with OA revealed significant efficacy in the WOMAC pain subscale score for each of the doses of fasinumab evaluated (1 mg, 3 mg, 6 mg, and 9 mg given every 4 weeks [Q4W]) compared with placebo (see current version of the Investigator's Brochure). Results from recent clinical studies with other anti-NGF antibodies, tanezumab (Pfizer) and fulranumab (Janssen), also support the role of NGF in pain modulation in patients with pain due to OA of the knee and hip (Brown 2012, Hefti 2006, Lane 2010) and in patients with chronic low back pain (Katz 2011, Kivitz 2013).

In all clinical studies completed to date, fasinumab was generally well tolerated. Arthralgia, joint swelling, peripheral edema, hypoesthesia, and myalgia were more frequently reported in fasinumab-treated patients than in placebo-treated patients. In neurological evaluations, abnormalities in vibration sense were more frequent in the fasinumab patients than in the placebo patients. These adverse events (AEs) or physical examination abnormalities associated with fasinumab were generally mild to moderate in intensity and were transient (see current version of the Investigator's Brochure).

Data from studies of tanezumab and fulranumab indicated that these molecules were associated with an increased risk of destructive arthropathy (DA), a unique clinical form of rapidly progressive arthropathy over and above that seen in the normal progression of osteoarthritis. Analyses of the tanezumab data by its sponsor, defined by anatomic pathological criteria on specimens obtained on joint replacement (JR), revealed that the risk of DA increases with tanezumab dose and is further increased with the concomitant use of chronic NSAIDs (>90 days) (Lane 2010). Most cases of DA occurred in joints with a documented history of OA.

Based on the potential risk of DA identified in tanezumab and fulranumab, the US Food and Drug Administration (FDA) placed the class of anti-NGF antibodies on clinical hold in 2010. Following a review of anti-NGF antibody clinical data in March 2012, the FDA determined that clinical studies of anti-NGF therapies could resume if mitigation strategies were implemented to minimize

the risk of DA. To address concerns about potential events of DA, a risk-mitigation approach is also being implemented for all fasinumab studies, as outlined in Section 9.6.1.1. This approach includes sensitive, prospective, and rigorous radiologic screening and monitoring for select changes in joint structure. Patients who develop these changes, which are referred to throughout this document as adjudicated arthropathy (AA), are required to discontinue study therapy.

Since the removal of the FDA clinical hold, Regeneron Pharmaceuticals, Inc, (Regeneron) has conducted or initiated several clinical studies of fasinumab. In all clinical studies to date, fasinumab was associated with a low rate of discontinuations due to AEs. Patients treated with fasinumab generally had more frequent events than did placebo-treated patients of arthralgia, joint swelling, peripheral edema, altered peripheral sensation (eg, paresthesia, dysesthesia), and myalgia.

In the phase 2/3 study of fasinumab in patients with pain due to OA of the knee or hip (R475-PN-1227), 26 AA events occurred in 24 patients. There was an increase in AA events that appeared to be related to greater fasinumab dose. Although these events were milder than the severe DA events presented at the 2012 FDA Arthritis Advisory Committee, in consideration of the lack of an observed dose response for efficacy in OA, the risk-benefit ratio was deemed unfavorable for the fasinumab 6 mg Q4W and 9 mg Q4W doses in patients with OA in comparison to the other fasinumab doses that were studied (ie, 1 mg Q4W and 3 mg Q4W). The dose regimens that were being evaluated in the phase 3 studies for OA pain in the knee or hip included 1 mg Q8W, 1 mg Q4W, 3 mg Q4W, and 6 mg Q8W. In April 2018, the independent Data Monitoring Committee (DMC) recommended discontinuing 6 mg Q8W and 3 mg Q4W (expected to have similar exposure to 6 mg Q8W) based on a review of unblinded data in study R475-PN-1523. Subsequently, a small Regeneron team reviewed the data and agreed with this recommendation. The DMC noted imbalances in clinically relevant AEs including time to total joint replacement, peripheral edema, arthralgia and a trend towards early fractures. The phase 3 program for OA pain in the hip or knee will continue to evaluate fasinumab 1 mg with the highest dose regimen of 1 mg Q4W, which is supported by the independent DMC as having a favorable benefit-risk profile.

In 2012, studies of other anti-NGF monoclonal antibodies identified adverse changes in the sympathetic nervous system (SNS) of mature animals of several species (rat and non-human primate). These effects included a reversible decrease in neuron volume. To date, no statistically significant or consistent effects of fasinumab on the SNS have been detected in animal studies with up to 6 months of treatment. Fasinumab has sub-picomolar affinity for human NGF (0.35pM). Fasinumab has little or no affinity for other neurotrophin family members, showing no detectable binding to either brain-derived neurotrophic factor (BDNF) or neurotrophin 3 (NT-3). At high concentrations, fasinumab shows low affinity binding to neurotrophin 4 (NT-4) (344nM).

Fasinumab's high specificity for NGF could potentially limit its nervous system impact relative to other anti-NGF antibodies with less specificity. Some populations of neurons, such as proprioceptive neurons and some visceral neurons, preferentially express TrkC as their neurotrophin receptor. The only neurotrophin that can activate TrkC is NT-3, so blocking NT-3 could compromise the integrity of these populations of neurons. NT-3 appears to have functional benefit in adult organisms. For instance, NT-3 has been shown to be neuroprotective for proprioceptive neurons using nerve conduction studies in adult rats (Liu 2011). NT-3 has also shown efficacy against constipation in adult patients, and is therefore thought to play a role in bowel motility (Parkman 2003). Based on the potential risk of SNS toxicity associated with other

anti-NGF monoclonal antibodies in animal studies, a risk mitigation approach is being implemented for all fasinumab studies, as outlined in Section 9.6.1.2.

Fasinumab is currently being evaluated in 3 ongoing phase 3 studies in OA patients. Study R475-PN-1523 is designed to assess the long-term safety and efficacy of multiple doses of fasinumab compared to placebo in patients with pain due to OA of the hip or knee. Study R475-OA-1611 is designed to compare the efficacy and safety of fasinumab to placebo and to naproxen, a standard-of-care NSAID for moderate-to-severe pain due to OA of the hip or knee. Study R475-OA-1688 is designed to compare the efficacy and safety of fasinumab to placebo, and to a pooled NSAID arm (celecoxib or diclofenac, which are additional standard-of-care NSAIDs for moderate-to-severe pain due to OA of the hip or knee).

The phase 2 study described here is designed to evaluate the neurological safety of fasinumab compared to placebo on nerve impulse transmission in motor and sensory nerves. Potential SNS symptoms will be monitored using the Survey of Autonomic Symptoms and through assessments of orthostatic hypotension.

Additional background information on the study drug and development program may be found in the current version of the Investigator's Brochure. A benefit-risk statement for fasinumab is also provided in the Investigator's Brochure.

### 2. STUDY OBJECTIVES

### 2.1. Primary Objective

The primary objective of the study is to evaluate the effect of fasinumab compared to placebo on peripheral nerves in patients with pain due to OA of the hip or knee.

### 2.2. Secondary Objectives

The secondary objectives of the study are:

- To evaluate the efficacy of fasinumab compared to placebo in patients with pain due to OA of the hip or knee
- To evaluate the safety and tolerability of fasinumab compared to placebo in patients with pain due to OA of the hip or knee
- To characterize the concentrations of fasinumab in serum in patients with pain due to OA of the hip or knee
- To evaluate the immunogenicity of fasinumab in patients with pain due to OA of the hip or knee

### 3. RATIONALE

### 3.1. Rationale

### 3.1.1. Rationale for Study Design

The present study is a randomized, double-blind, placebo-controlled, multicenter study to evaluate the neurological safety and efficacy of fasinumab in patients with OA of the knee or hip who have a history of inadequate pain relief for their OA pain from acetaminophen/paracetamol, and a history of intolerance to or inadequate pain relief from oral NSAIDS and opioids (or are unwilling to take opioids) for OA pain management. This study will evaluate the neurological safety of fasinumab compared to placebo in OA patients treated for up to 16 weeks by measuring nerve conduction velocities and evoked amplitudes of the peroneal, ulnar, and sural nerves. This study will also provide additional safety, tolerability, efficacy, pharmacokinetic (PK), and immunogenicity data for fasinumab.

The target study population was chosen because they currently have unmet medical needs with respect to unacceptable pain control, in spite of the availability of current analgesic treatment options. The study will be conducted with appropriate eligibility criteria to exclude patients who may be at risk for events of joint damage and SNS effects. Furthermore, specific questionnaires and physical examinations will be employed to monitor for any events of arthralgia, worsening joint pain, altered peripheral sensation, AA, and SNS effects. All patients included in the study will have regular study visits and receive diagnostic procedures (ie, X-rays, magnetic resonance imaging [MRI]) to evaluate their ongoing OA. Adverse event monitoring will be ongoing throughout the trial.

The inclusion of a placebo treatment group is important to accurately determine the neurological safety, overall safety, and efficacy of fasinumab and to more accurately estimate the risk of AEs, including the adverse events of special interest (AESI) of AA, SNS dysfunction, and altered peripheral sensation. Rescue medication (paracetamol/acetaminophen) will be made available for any patient with breakthrough pain. Therefore, the use of a placebo group is justified, as placebo-treated patients will not be placed at significant risk. Patients and investigators can choose to end participation at any time.

The patients will be stratified by the affected index joint (hip or knee) and by Kellgren-Lawrence (K-L) score (2 to 3, or 4) of the index joint at screening to enable analysis of efficacy and safety. The use of a K-L stratification scheme ensures that there is an equal distribution of patients with the most severe OA at baseline across the treatment groups.

#### 3.1.2. Rationale for Dose Selection

In this study, patients will be randomized to receive fixed-dose, subcutaneous (SC) injections of 1 mg fasinumab Q4W or placebo Q4W. The 1 mg Q4W dose regimen is the highest dose regimen (exposure) under evaluation in the fasinumab phase 3 OA pain program. This dose regimen is anticipated to have a favorable benefit-risk profile in patients with OA pain.

### 4. STUDY VARIABLES

### 4.1. Demographic and Baseline Characteristics

Baseline characteristics will include standard demography (eg, age, race, weight, height, etc.), disease characteristics including medical and surgical history, and medication history for each patient.

### 4.2. Primary and Secondary Endpoints

### 4.2.1. Primary Endpoints

The primary endpoints of the study are:

- Change from baseline to week 16 in peroneal motor nerve conduction velocity
- Change from baseline to week 16 in peroneal motor nerve action potential amplitude
- Change from baseline to week 16 in sural sensory nerve conduction velocity
- Change from baseline to week 16 in sural sensory nerve action potential amplitude
- Change from baseline to week 16 in ulnar sensory nerve conduction velocity
- Change from baseline to week 16 in ulnar sensory nerve action potential amplitude

### 4.2.2. Secondary Endpoints

The secondary endpoints of the study are:

- Change from baseline to week 16 in WOMAC pain subscale score
- Change from baseline to week 16 in WOMAC physical function subscale score

### 4.3. Additional Safety Endpoints

Additional safety endpoints in this study include:

- Incidence of AA (as confirmed by an independent adjudication committee) through week 36
- Incidence of DA (as confirmed by an independent adjudication committee) through week 36
- Incidence of treatment-emergent adverse event (TEAEs) through week 16
- Incidence of SNS dysfunction (as diagnosed after consultation with an appropriate specialist, such as a neurologist and/or cardiologist) through week 36
- Incidence of peripheral sensory AEs that require a neurology or other specialty consultation through week 36
- Incidence of all-cause joint replacement (JR) surgeries week 36
- Incidence of JRs at telephone survey approximately 52 weeks after last dose of study drug

#### 4.4. Pharmacokinetic Variables

The PK variable is the concentration of functional fasinumab in serum samples collected at each time point. Samples in this study will be collected using a sparse sampling schedule. These sampling time points are specified in Table 1.

### 4.5. Anti-Drug Antibody Variables

Anti-drug antibody (ADA) variables include status (positive or negative), titer, and time point/visit. Samples in this study will be collected at the visits specified in Table 1.

### 5. STUDY DESIGN

### 5.1. Study Description and Duration

This is a phase 2, randomized, double-blind, placebo-controlled, multicenter study designed to evaluate the neurological safety of fasinumab compared to placebo in patients with pain due to OA of the hip or knee.

The study duration will be approximately 64 weeks starting at randomization (day 1). The study consists of a screening period of up to 30 days, a 7- to 10-day pre-randomization period (7 days with a +3 day window), a 16-week treatment period (with the last Q4W dose of study drug administered at week 12), a 20-week follow-up period, and a final phone contact approximately 52 weeks after the last dose of study drug is administered (Figure 1).

Figure 1: Study Flow Diagram



EOS- End of study

### 5.1.1. Screening and Pre-Randomization

Prior to randomization, patients will undergo screening procedures, including X-ray of the shoulders, hips, and knees. Magnetic resonance imaging of the index and contralateral joints must be performed at screening and the results assessed by the central imaging vendor. In addition, an MRI will be performed on any knee or hip joint with a K-L score of  $\geq 3$ . Randomization visits cannot occur until there is confirmation from the central imaging vendor that there are no exclusionary findings on the X-rays and any required MRIs.

Prior to randomization, patients will also undergo nerve conduction assessments. Patients must complete all other inclusion/exclusion assessments before undergoing the nerve conduction

assessments. Randomization cannot occur until there is confirmation from the central reader assessment that the results are within the established parameters.

During the screening period, patients may continue to take their current treatment regimen for OA pain.

Patients eligible for the study will complete a pre-randomization period, during which all pain medication, except for the study-provided rescue medication (acetaminophen/paracetamol), will be discontinued. The pre-randomization visit will be 7 to 10 days (7 days with a +3 day window) before the randomization visit. Patients will discontinue and/or undergo a washout of their current pain medications for OA during the pre-randomization period. As needed, during this pre-randomization period, patients may take acetaminophen/paracetamol for pain relief according to the regional standard-of-care (see Section 7.2 for details). Acetaminophen/paracetamol must not be taken within 24 hours prior to the randomization visit.

### 5.1.2. Rescreening

### Retesting during the Screening and Pre-Randomization Periods

An assessment that fails to meet eligibility criteria may be repeated once within the screening or pre-randomization period when approved by the sponsor or designated Medical Monitor under either of the following conditions: 1) The failure is believed by the investigator to be due to a condition that would resolve or could be treated; or 2) A laboratory value that minimally exceeds the cut-off value and is not clinically relevant. Only the assessments that did not meet the eligibility criteria require repetition, if done within the screening period or pre-randomization period. Patients may not repeat any assessments if they did not meet the WOMAC criteria, if they had orthostatic hypotension (defined in Section 8.2.3.4), or if the nerve conduction test showed results not within the established parameters as per central reader assessment during the screening or pre-randomization visit.

### Rescreening after Screen Failure

Rescreening can be completed for patients who fail to meet the screening visit window requirements or who are unable to complete all imaging assessments within the specified screening period. Patients who are rescreened after the pre-randomization window must be declared screen failures, be registered in the interactive web response system (IWRS) as a new patient with a new identification number, and then repeat all screening procedures, with the exception of imaging assessments. Any imaging assessments would need to be repeated only if they were taken more than 60 days from completion of the previous screening X-rays and MRI assessments. Patients cannot rescreen if they have screen failed due to not meeting the WOMAC criteria, if they have orthostatic hypotension (defined in Section 8.2.3.4), or if the nerve conduction test showed results not within the established parameters as per central reader assessment during the screening or prerandomization visit.

**R475-OA-1758 Amendment 2** 

#### 5.1.3. Randomization

On day 1 (baseline), approximately 180 patients will be randomized in a 1:1 ratio to the following treatment groups:

- Fasinumab 1 mg SC Q4W
- Fasinumab-matching placebo SC Q4W

Patients will receive treatment as described in Section 7.1. Randomization will be stratified according to the affected index joint (hip or knee) and the K-L score (2 to 3, or 4) at the screening visit.

#### **5.1.4.** Treatment Period

During the treatment period (day 1 through week 16), patients will be permitted to use only study-provided acetaminophen/paracetamol as rescue medication. Patients will record their use of acetaminophen/paracetamol in a diary. Patients should discontinue use of acetaminophen/paracetamol at least 24 hours prior to the start of each study visit in order to minimize the confounding effects of the rescue medication on efficacy measurements.

Neurological, efficacy, and safety assessments will be performed during the treatment period, as outlined in Table 1.

If a patient must undergo JR surgery during the treatment period, he or she will be asked to complete pre-operative imaging and to undergo post-surgery follow-up, as outlined in Table 2.

### **5.1.5.** Follow-up Period

Follow-up of patients will continue for an additional 20 weeks after the last treatment period visit. Patients will have 2 study visits during the follow-up period (week 26 and week 36). Neurological, efficacy and safety assessments will be performed during the follow-up period, as outlined in Table 1.

Patients will be directed not to take concomitant medications that contain NSAIDs (oral or topical, except up to 150 mg/day of aspirin, which is permitted for cardiac prophylaxis) until at least 16 weeks after the last study drug injection.

If a patient must undergo JR surgery during the follow-up period, he or she will be asked to complete pre-operative imaging and to undergo post-surgery follow-up, as outlined in Table 2.

### 5.1.6. End of Study Phone Contact and Additional Imaging

Phone contact will be made approximately 52 weeks after administration of the last dose of fasinumab or placebo to document patient status with regard to JR surgery (if patient underwent, is scheduled for, or is on a wait list for JR surgery). Additionally, patients who had an AA confirmed during the study will have an MRI performed of the AA joint(s). If the AA joint(s) have undergone JR, an X-ray may be substituted for an MRI.

#### **5.1.7.** Study Stopping Rules

An independent Data Monitoring Committee (DMC) will monitor unblinded data on an ongoing basis to assess the risk/benefit profile of fasinumab. Based on these reviews, in the context of the

totality of evidence, if the DMC has significant concerns at any time regarding a meaningful imbalance between treatment groups in joint-related AEs, SNS dysfunction, neurosensory disturbances, or any other safety issues, the DMC may make a recommendation to temporarily halt, alter, or terminate:

- individual dose groups within the study or across studies
- the full study (screening, randomization, dosing of study drug)
- the fasinumab program

for additional review and communication to regulatory authorities. Based on the outcome of the review and discussions with the appropriate regulatory authorities, the study may be suspended, restarted, or terminated.

Formal program wide statistical study stopping criteria for clinical studies involving fasinumab may be added to the DMC charter as deemed necessary by the sponsor, DMC and/or Health Authorities.

#### **5.1.8.** End of Study Definition

The end of study is defined as the last phone contact of the last patient in this study.

### **5.2.** Planned Interim Analysis

An interim analysis may be performed in order to provide peripheral nerve safety data for regulatory purposes.

### **5.3.** Study Committees

### **5.3.1.** Independent Data Monitoring Committee

An independent DMC will meet periodically to review unblinded data as the study progresses, and based on the findings, will make recommendations to the sponsors about the conduct of the study. The DMC will comprise independent statistical and medical experts. Further details will be defined in the DMC charter. Additional safety monitoring will occur on an ongoing basis by the Regeneron Safety Team.

### **5.3.2.** Arthropathy Adjudication Committee

An independent, expert, blinded adjudication committee composed of radiologists trained in musculoskeletal imaging will adjudicate all potential joint AEs of AA (defined in Section 9.6.1.1) as well as pre-operative images in patients undergoing JR.

# 6. SELECTION, WITHDRAWAL, AND REPLACEMENT OF PATIENTS

#### 6.1. Number of Patients Planned

The study will enroll approximately 180 patients at about 30 global sites. Each treatment group (fasinumab and fasinumab-matching placebo) will enroll approximately 90 patients.

### **6.2.** Study Population

Eligible patients for this study consist of men and women who are at least 18 years of age at the time of study entry with a clinical diagnosis at the screening visit of OA of the knee or hip, based on the American College of Rheumatology criteria, and with radiologic evidence of OA (K-L score  $\geq$ 2) at the index joint.

### **6.2.1.** Inclusion Criteria

A patient must meet the following criteria to be eligible for inclusion in the study:

- 1. Male and female patients ≥18 years of age at screening visit
- 2. Provide signed informed consent signed by study patient or legally acceptable representative
- 3. Body mass index ≤39 at screening visit
- 4. A clinical diagnosis of OA of the knee or hip based on the American College of Rheumatology criteria with radiologic evidence of OA (K-L score ≥2 for the index joint) at the screening visit, with the following definitions:
  - The index joint is defined as the joint with OA under evaluation for this study
  - A joint previously treated with JR surgery cannot be the index joint
  - A joint previously surgically modified within the past year cannot be the index joint (with the exception of cruciate ligament reconstruction surgery, patellar fracture repair surgery, or meniscal repair)
  - If a patient has a K-L score of ≥2 at more than 1 knee or hip joint, the index joint is the joint with the greatest WOMAC pain subscore at the screening visit
  - If 2 or more knee or hip joints have a K-L score of  $\geq$ 2 and the same WOMAC pain subscore, the index joint is the joint with the greater K-L score
  - If 2 or more joints have a K-L score of ≥2, the same WOMAC pain subscores, and the same K-L scores, then the investigator may choose 1 of these joints as the index joint
- 5. Moderate-to-severe pain in the index joint defined as a WOMAC average pain subscale score of  $\geq 4$  at both the screening and randomization visits
- 6. Willing to discontinue current pain medications and to adhere to study requirements for rescue treatments (paracetamol/acetaminophen to be taken as needed with a maximum daily dose of 2500 mg [countries where 500 mg strength tablets/capsules are available] or 2600 mg [countries where 325 mg strength tablets/capsules are available])
- 7. A history of at least 12 weeks of analgesics use for pain due to OA of the knee or hip, as defined by:
  - a. Inadequate pain relief from acetaminophen/paracetamol AND
  - b. Intolerance to or inadequate pain relief from at least 1 oral NSAID AND

- c. Intolerance to or inadequate pain relief from opioid or tramadol therapy, unwillingness to take opioid or tramadol therapy for a medically acceptable reason, or lack of access to an opioid or to tramadol
- 8. A history of regular use of analgesic medications for OA pain (defined as an average of 4 days per week over the 4 weeks prior to the screening visit), including oral NSAIDs, selective cyclooxygenase 2 inhibitors, opioids, paracetamol/acetaminophen, or combinations thereof
- 9. Consent to allow all radiographs and medical/surgical/hospitalization records of care received elsewhere prior to and during the study period to be shared with the investigator
- 10. Willing to maintain current activity and exercise levels throughout the study
- 11. Willing and able to comply with clinic visits and study-related procedures and willing to provide follow-up information related to any JR surgery that occurs within the period of time covered by their intended participation in the study
- 12. Able to understand and complete study-related questionnaires

#### **6.2.2.** Exclusion Criteria

A patient who meets any of the following criteria will be excluded from the study:

- 1. History or presence at the screening visit of non-OA inflammatory joint disease (eg, rheumatoid arthritis, lupus erythematosus, psoriatic arthritis, pseudo-gout, gout, spondyloarthropathy, polymyalgia rheumatica, joint infections within the past 5 years), Paget's disease of the spine, pelvis or femur, neuropathic disorders, multiple sclerosis, fibromyalgia, tumors or infections of the spinal cord, or renal osteodystrophy
- 2. History or presence on imaging of arthropathy (osteonecrosis, subchondral insufficiency fracture, rapidly progressive OA type 1 or type 2), stress fracture, recent stress fracture, neuropathic joint arthropathy, hip dislocation (prosthetic hip dislocation is eligible), knee dislocation (patella dislocation is eligible), congenital hip dysplasia with degenerative joint disease, extensive subchondral cysts, evidence of bone fragmentation or collapse, or primary metastatic tumor with the exception of chondromas or pathologic fractures during the screening period
- 3. Trauma to the index joint within 3 months prior to the screening visit
- 4. History or presence of signs or symptoms of compression neuropathy, including carpal tunnel syndrome or sciatica
- 5. Patient is not a candidate for MRI
- 6. Is scheduled for a JR surgery to be performed during the study period or who would be unwilling or unable to undergo JR surgery if one eventually became necessary
- 7. Patients with nerve conduction results (for the peroneal, sural, and ulnar nerves) that are outside of the established parameters, based on standards detailed in the study manual and according to the eligibility report provided by the central reader

- 8. Patients receiving, or who plan to receive, interventions, devices, or medications that alter nerve conduction or are contraindicated in patients undergoing nerve conduction studies (eg, edema, tarsal tunnel syndrome)
- 9. History or presence at the screening visit of autonomic neuropathy, diabetic neuropathy, or other peripheral neuropathy, including reflex sympathetic dystrophy and complex regional pain syndrome
- 10. History or diagnosis of chronic autonomic failure syndrome including pure autonomic failure, multiple system atrophy (Shy-Drager syndrome)
- 11. Known allergy or sensitivity to monoclonal antibodies
- 12. Poorly controlled diabetes (defined as any single value of hemoglobin A1c [HbA1c] >9.0%) at the screening visit
- 13. Known history of human immunodeficiency virus (HIV) infection
- 14. Known history of ocular herpes simplex virus, herpes simplex virus pneumonia, or herpes simplex virus encephalitis
- 15. History of sickle cell disease, including sickle cell anemia and β-thalassemia
- 16. Confirmed elevated screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2.5 times the upper limit of normal (ULN)
- 17. Resting heart rate of <50 beats per minute (bpm) or >100 bpm (by vital sign assessment or as captured during electrocardiogram [ECG] assessment) at the screening or randomization visits
- 18. History or presence of 2<sup>nd</sup> or 3<sup>rd</sup> degree heart block, 1<sup>st</sup> degree heart block with abnormal QRS complex, or bifascicular block by ECG assessment at the screening visit
- 19. History or presence of orthostatic hypotension, as defined in Section 8.2.3.4, at the screening, pre-randomization, or randomization visits
- 20. History of poorly controlled hypertension, as defined by:
  - a. Systolic blood pressure ≥180 mm Hg or diastolic blood pressure ≥110 mm Hg at the screening visit
  - b. Systolic blood pressure of 160 mm Hg to 179 mm Hg or diastolic blood pressure of 100 mm Hg to 109 mm Hg at the screening visit, AND a history of end-organ damage (including history of left ventricular hypertrophy, heart failure, angina, myocardial infraction, stroke, transient ischemic attack, peripheral arterial disease and moderate to advanced retinopathy [hemorrhages or exudates, papilledema])
- 21. Congestive heart failure with New York Heart Classification of stage III or IV (Dolgin 1994)
- 22. Transient ischemic attack or cerebrovascular accident within the past 12 months prior to the screening visit, or myocardial infarction, or acute coronary syndromes within the past 6 months prior to the screening visit

- 23. Significant concomitant illness including, but not limited to, psychiatric, cardiac, renal, hepatic, neurological, endocrinological, metabolic, or lymphatic disease that, in the opinion of the investigator, would adversely affect the patient's participation in the study
- 24. New major illness diagnosed within 2 months prior to the screening visit
- 25. Known history of infection with hepatitis B virus. Patients with a history of hepatitis B are eligible if there is documentation of a negative test for hepatitis B surface antigen and a positive test for antibodies to the hepatitis B virus surface antigen
- 26. Known history of infection with the hepatitis C virus. Patients with a history of hepatitis C are eligible if there is documentation of a negative hepatitis C virus RNA test
- 27. History or presence of malignancy within the last 5 years prior to screening, except patients who have been treated successfully with no recurrence for >1 year of basal cell or squamous cell carcinoma of the skin or in-situ cervical cancer
- 28. History of hospital admission for depression or suicide attempt within 5 years or active, severe major depression at screening
- 29. Use of systemic (ie, oral or intramuscular) corticosteroid within 30 days prior to the screening visit. Intra-articular corticosteroids in the index joint within 12 weeks prior to the screening visit, or to any other joint within 30 days prior to the screening visit (topical, intra-nasal, and inhaled corticosteroids are permitted)
- 30. Use of a monoamine reuptake inhibitor, tricyclic antidepressants, selective serotonin reuptake inhibitors and serotonin norepinephrine reuptake inhibitors for treatment of pain within 4 weeks prior to the screening visit
- 31. Has positive urine drug test results during screening (eg, amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates), unless in the opinion of the investigator, the positive test results may be due to the patient's current permitted medications
- 32. History of (within 5 years prior to the screening visit) or current alcoholism, alcohol abuse, substance abuse, or abuse of prescription pain medication
- 33. History of cannabis use for the treatment of pain within the past 6 months prior to the screening visit
- 34. Ongoing participation in a clinical research study evaluating another investigational drug or having received another investigational product within 30 days or 5 half-lives of the screening visit, whichever is longer
- 35. Exposure to an anti-NGF antibody prior to the screening visit or known sensitivity or intolerance to anti-NGF antibodies or participation in a clinical trial evaluating anti-NGF antibodies
- 36. Member of the clinical site study team and/or his/her immediate family, unless prior approval granted by the sponsor
- 37. Pregnant or breastfeeding women

- 38. Women of childbearing potential who have a positive pregnancy test result or do not have their pregnancy test result at baseline
- 39. Women of childbearing potential\* who are unwilling to practice highly effective contraception prior to start of the first treatment, during the study, and for at least 20 weeks after the last dose. Highly effective contraceptive measures include:
  - a. stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening
  - b. intrauterine device (IUD); intrauterine hormone-releasing system (IUS)
  - c. bilateral tubal ligation
  - d. vasectomized partner
  - e. and or sexual abstinence<sup>†‡</sup>
- \* Postmenopausal women must be amenorrheic for at least 12 months (without an alternative medical cause) in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented complete hysterectomy or tubal ligation.
- † Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.
- ‡ Periodic abstinence (calendar, symptothermal, and post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method (LAM) are not acceptable methods of contraception. Female condom and male condom should not be used together.

Note: HIV and/or hepatitis testing will be performed on a country-by-country basis, according to local guidelines if required by regulatory authorities or ethics boards.

### 6.3. Premature Withdrawal from the Study

A patient has the right to withdraw from the study at any time, for any reason, and without repercussion.

The investigator and/or sponsor have the right to withdraw a patient from the study if it is no longer in the interest of the patient to continue in the study, or if the patient's continuation in the study places the scientific outcome of the study at risk (eg, if a patient does not or cannot follow study procedures). An excessive rate of withdrawals would render the study uninterpretable; therefore, unnecessary withdrawal of patients should be avoided.

Patients who are withdrawn prematurely from the study will be asked to complete the early termination visit, as described in Section 8.1.3.

Rules for discontinuation of study treatment (permanent or temporary) are discussed in Section 7.3.2.

### **6.4.** Replacement of Patients

Patients prematurely withdrawn from the study or study drug will not be replaced.

#### 7. STUDY TREATMENTS

### 7.1. Investigational and Reference Treatments

Fasinumab drug product is supplied for this study in the following concentrations:

- Fasinumab 2 mg/mL: Each 1 mL single-use pre-filled syringe delivers 0.5 mL of 2 mg/mL solution to provide a 1 mg dose of study drug
- Fasinumab-matching placebo: Each 1 mL single use pre-filled syringe delivers 0.5 mL of placebo solution.

All patients will receive SC injections of fasinumab or fasinumab-matching placebo. Patients will be randomized to 2 treatment groups in a 1:1 ratio to receive either fasinumab 1 mg SC Q4W or fasinumab-matching placebo SC Q4W. All SC injections will be in the abdomen, thigh, or upper arm. Instructions for dose preparation and study drug administration are provided in the pharmacy manual. Patients will be observed in the clinic for approximately 1 hour after study drug is administered.

Doses of study drug must be given within  $\pm 7$  days from the scheduled dose date. If the window is missed, the dose should not be administered. The next dose should be administered at the next scheduled dosing date.

### 7.2. Rescue Treatment

Starting at pre-randomization to the end of the 16-week treatment period, study-provided acetaminophen/paracetamol is the only allowed rescue medication. In the event of inadequate pain relief for OA or in the event of other pain (eg, headache) or fever, 1 to 2 tablets/capsules of study-provided acetaminophen/paracetamol may be taken no less than 4 hours apart as needed according to the local standard of care. The maximum allowed daily dose during the treatment and follow up periods is 2500 mg (500 mg x 5 tablets/capsules) in countries where 500 mg strength tablets/capsules are available or 2600 mg (325 mg x 8 tablets/capsules) in countries where 325 mg strength tablets/capsules are available (eg, North America). Where 500 mg strength tablets/capsules are available, the highest individual single dose is 1 gram. Where 325 mg tablets/capsules are available, the highest individual single dose is 650 mg.

In order to prevent severe liver damage, patients should be cautioned to avoid consumption of alcoholic beverages while on paracetamol/acetaminophen. Patients should also be cautioned not to take rescue medication at intervals of fewer than 4 hours and to take no more than the maximum allowable single dose (1 to 2 tablets/capsules) or maximum allowable total daily dose.

Acetaminophen/paracetamol must not be taken within 24 hours prior to scheduled study visits during the treatment period in order to minimize the confounding effects of rescue medication on efficacy assessment measures. Use of acetaminophen/paracetamol as study-provided rescue medication during the treatment period will be reported daily using diaries.

Acetaminophen/paracetamol accountability will be conducted at each study site visit starting at the baseline visit and continuing through the week 16 visit.

During the treatment period, acetaminophen/paracetamol will be sourced by the study sites and reimbursed by the sponsor unless country-specific regulations and customs require a different approach.

During the 20-week follow-up period, if acetaminophen/paracetamol is used, dosing instructions will be the same as during the treatment period including the maximum allowed daily dose. Use of acetaminophen/paracetamol will be captured as a concomitant medication during the follow-up period.

### 7.3. Dose Modification and Study Treatment Discontinuation Rules

#### 7.3.1. Dose Modification

Study drug dose modification for an individual patient is not allowed.

### 7.3.2. Study Drug Discontinuation

Study drug may be temporarily or permanently discontinued due to medical need, as determined by the investigator, medical monitor, or the sponsor and according to the study stopping rules (Section 5.1.7).

Patients who permanently discontinue from study drug will be encouraged to remain in the study and to complete all study assessments. Patients who agree and thus <u>do not withdraw from the study</u> will be asked to return to the clinic for all remaining study visits per Table 1.

Patients who permanently discontinue from study drug and who opt to withdraw from the study will be asked to complete an early termination visit (Section 8.1.3).

Patients who discontinue from study drug prior to study completion due to an AA (see Section 9.6.1.1) should return to the clinic for all remaining study visits per the visit schedule.

In the event that a patient must undergo JR surgery during the treatment or follow-up periods, he/she will be discontinued from study drug and asked to return to the study site for a pre-operative visit and for follow-up safety evaluations 4 and 20 weeks after surgery (as described in Section 8.2.4.7). Pre-operative imaging (X-rays and/or MRI) will be obtained and submitted to the independent adjudication committee for review to exclude or confirm the presence of an AA event. Instructions for the submission process are provided in the study manual.

### 7.3.2.1. Reasons for Permanent Discontinuation of Study Drug

Study drug dosing will be permanently stopped in the event of:

- A patient developing clinically significant peripheral sensory or motor neurologic events confirmed by a neurologist's examination and graded by the neurologist as at least moderate peripheral neuropathy limiting activities of daily living, ie, grade ≥2 according to Common Terminology Criteria for Adverse Events (CTCAE) v.4; study sites should use CTCAE v.4 criteria throughout the study for consistency
- Evidence of pregnancy
- A patient developing signs and symptoms indicative of carpal tunnel syndrome
- Continued noncompliance with protocol-defined maximum acetaminophen/ paracetamol use (with a maximum daily dose of 2500 mg [countries where 500 mg strength tablets/capsules are available] or 2600 mg [countries where 325 mg strength tablets/capsules are available]) during the treatment and follow-up periods, after appropriate counseling
- Continued noncompliance with the protocol, including usage of NSAIDs or other medications or non-pharmacologic treatments that are not permitted in the study, after appropriate counseling
- JR surgery
- AESI:
  - Adjudicated arthropathy, as described in Section 9.6.1.1.
  - Sympathetic nervous system dysfunction, as described in Section 9.6.1.2.
- Per protocol repeated nerve conduction test that confirms results are not within the established parameters for peroneal, sural, or ulnar nerves, as per central reader assessment and the neurologist's evaluation that confirms the diagnosis of peripheral neuropathy.
- Hepatotoxicity. Study drug should be discontinued if the following are observed:
  - 1. Total bilirubin (TBL) >2x ULN or international normalized ratio (INR) >1.5, and
  - 2. ALT or AST >3x ULN, and
  - 3. No other cause for 1 and 2 is readily apparent

Other causes of ALT, AST, and TBL elevations may include alcoholic hepatitis, autoimmune hepatitis, non-alcoholic hepatitis, heritable diseases (Gilbert's Syndrome), heart failure, and viral hepatitis.

NOTE: Study drug may be withheld in patients who do not meet criteria for permanently discontinuing study drug, until an alternative cause for drug-induced liver injury can be determined. The patient may be re-challenged if an alternative cause for elevated liver function tests is found and the liver function tests return to baseline, but only after discussion with the sponsor.

- Systemic hypersensitivity reaction deemed by the investigator to be related to study drug
- Any other medical need, as determined by the investigator
- Sponsor decision
- Patient withdraws consent

## 7.3.2.2. Reasons for Temporary Discontinuation of Study Drug

Study drug may be temporarily discontinued due to medical need, as determined by the investigator. Study drug will be temporarily withheld while awaiting imaging adjudication for worsening joint pain or when routine imaging suggests AA and prompts the need for additional imaging (see Section 9.6.1.1), for patients who are determined to have orthostatic hypotension or determined to have new or worsening symptoms suggestive of SNS dysfunction while awaiting evaluation by a specialist (see Section 9.6.1.2), or for patients with symptoms of peripheral neuropathy while awaiting evaluation by a specialist and/or results of a nerve conduction test (see Section 9.6.1.3).

Study drug should not be re-started until the next study visit, unless imaging, nerve conduction test results, or neurology evaluation results are available within the current visit window and confirm that study drug may be restarted.

## 7.4. Management of Acute Reactions

## 7.4.1. Systemic Injection Reactions

Emergency equipment and medication for the treatment of systemic reactions must be available for immediate use. All systemic injection reactions must be reported as AEs (as defined in Section 9.3.1) and graded using the grading scales as instructed in Section 9.5.1.

Acute systemic reactions following SC injection of study drug should be treated using clinical judgment to determine the appropriate response according to typical clinical practice.

## 7.4.2. Local Injection Site Reactions

Local injection site reactions must be reported as AEs and graded according to Section 9.5.1.

# 7.5. Method of Treatment Assignment

Approximately 180 patients will be randomized in a 1:1 ratio to receive fasinumab (1 mg SC Q4W) or fasinumab-matching placebo (Q4W) according to a central randomization scheme provided by an IWRS to the designated study pharmacist (or qualified designee). Randomization will be stratified according to the affected index joint (hip or knee) and the K-L score (2 to 3, or 4) at the screening visit.

## 7.5.1. Blinding

Study patients, the principal investigators, and study site personnel will remain blinded to all randomization assignments throughout the study. The Regeneron study team and contract research organization (CRO) personnel who are in regular contact with the study site will remain blinded to all patient randomization assignments.

Blinded study drug kits coded with a drug numbering system will be used. In order to maintain the blind, lists linking these codes with product lot numbers will not be accessible to individuals involved in study conduct.

Anti-drug antibody results will not be communicated to the sites before the end of the study, and the sponsor operational team will not have access to results associated with patient identification until after the final database lock.

Selected individuals not involved in the conduct of the study may have access to unblinded data as needed for safety review or other data review. No study personnel involved in the day-to-day conduct of the study will have access to unblinded data before the database is locked for this study.

## 7.5.2. Emergency Unblinding

Unblinding of treatment assignment for a patient may be necessary due to a medical emergency or any other significant medical event (eg, pregnancy).

If unblinding is required:

- Only the investigator will make the decision to unblind the treatment assignment
- Only the affected patients will be unblinded
- The designated study pharmacist(s)/designee at the study site will provide the treatment assignment to the investigator. If there is no study pharmacist, the investigator for the site will unblind the patient
- The investigator will notify Regeneron and/or designee as soon as possible after unblinding the patient

Treatment assignment is not to be provided to site personnel, other than the unblinded study pharmacist (when applicable), at any time during the conduct of the study, except in the case of a true emergency. In the event that there is no study pharmacist, the individual at the site fulfilling that role will be the only unblinded member of the site personnel.

## 7.5.3. Unblinding for Regulatory Reporting Purposes

Treatment assignments for certain patients may be unblinded to Pharmacovigilance and Risk Management personnel for the purpose of regulatory reporting of Suspected Unexpected Serious Adverse Reactions (SUSARs).

# 7.6. Treatment Logistics and Accountability

## 7.6.1. Packaging, Labeling, and Storage

A medication numbering system will be used to label blinded investigational study drug. Lists linking medication numbers with product lot numbers will be maintained by the groups (or companies) responsible for study drug packaging. In order to maintain the blind, these lists will not be accessible to individuals involved in study conduct.

Study drug will be stored at the site at a temperature of 2°C to 8°C. Storage instructions will be provided in the pharmacy manual.

## 7.6.2. Supply and Disposition of Treatments

Study drug will be shipped at a temperature of 2°C to 8°C to the investigator or designee at regular intervals or as needed during the study. At specified time points during the study (eg, interim site

monitoring visits), at the site close-out visit, and following drug reconciliation and documentation by the site monitor, all used drug will be destroyed at site while unused drug will be returned to the sponsor or designee. Refer to pharmacy manual for details.

## 7.6.3. Treatment Accountability

All drug accountability records must be kept current.

The investigator must be able to account for all used and unused study drug. These records should contain the dates, quantity, and study drug that is:

- dispensed to each patient,
- returned from each patient (if applicable),
- disposed of at the site, or returned to the sponsor or designee.

All accountability records must be made available for inspection by the sponsor and regulatory agency inspectors; photocopies must be provided to the sponsor at the conclusion of the study.

## 7.6.4. Treatment Compliance

All study drug compliance records must be kept current and made available for inspection by the sponsor and regulatory agency inspectors.

## 7.7. Concomitant Medications and Procedures

Any treatment administered and/or procedures performed from screening to the end of the follow-up period will be considered concomitant medication and/or procedures, respectively. This includes medications and/or procedures that were started before the study and are ongoing during the study.

#### 7.7.1. Prohibited Medications

Patients will be required to discontinue all non-study pain medication (oral or topical; except up to 150 mg/day of aspirin/aminosalicylic acid [5-ASA], which is permitted for cardiac prophylaxis, per local guidelines), starting at the pre-randomization visit and through the treatment period.

Opioid analgesic medications (including tramadol) are prohibited through the week 16 study visit. Patients will be directed not to take concomitant medications that contain NSAIDs (oral or topical, except up to 150 mg/day of aspirin, which is permitted for cardiac prophylaxis) until at least 16 weeks after the last study drug injection. A list of medications containing NSAIDs will be provided in the study reference manual and in a reference card given to patients.

Other excluded medications during the treatment period include:

- Any other investigational agent
- Medical or regular recreational use of marijuana
- Chondroitin sulfate
- Glucosamine
- Hyaluronic Acid Intra-articular Injections

- Muscle relaxants including cyclobenzaprine, carisoprodol, orphenadrine, tizanidine (see Section 7.7.2 for permitted muscle relaxants)
- Corticosteroids (topical, intranasal, and inhaled formulations are permitted), adrenocorticotropic hormone
- Cyclosporine, methotrexate, mycophenolate mofetil, tacrolimus
- Azathioprine, sulfasalazine, hydroxychloroquine
- IL-6 or IL-6 receptor antagonists
- Abatacept, ustekinumab
- Tumor necrosis factor antagonists
- IL-1 inhibitors, including diacerein
- Apremilast, and tofacitinib

#### 7.7.2. Permitted Medications and Procedures

Patients receiving chronic medication therapy must be on a stable dose of such medication for at least the 30 days prior to the screening visit. Monoamine reuptake inhibitors, tricyclic antidepressants, selective serotonin reuptake inhibitors, and serotonin norepinephrine reuptake inhibitors are permitted for non-pain-related treatment. Patients must be on therapy for at least 8 consecutive weeks and on a stable dose for at least 4 weeks prior to the screening visit and throughout the planned duration of the patient's participation in the study.

Low-dose aspirin/5-ASA (up to 150 mg/day) for cardiac prophylaxis is permitted. Acetaminophen/paracetamol taken acutely for treatment of non-OA pain is permitted, however, the total daily dosage limits cannot be exceeded regardless of the reason for acetaminophen/paracetamol use. During the pre-randomization and treatment periods, acetaminophen/paracetamol use will be captured in the diary; use for relief of pain other than pain due to OA will be reported in the diary as "other". During the screening and follow-up periods, acetaminophen/paracetamol taken for any reason should be reported as concomitant medication. Topical steroids are permitted.

Muscle relaxants, such as Skelaxin® (metaxalone) and others, are permitted. Prohibited muscle relaxants are listed in Section 7.7.1.

Physical therapies (such as transcutaneous electrical nerve stimulation and acupuncture) are permitted during the trial, provided that patients have been on a stable regimen for at least 4 weeks prior to entering into the trial and that they expect to maintain this regimen during the trial.

Joint replacement is a permitted procedure during the study (see Section 8.2.4.7 for procedures to be followed in the event of JR).

## 8. STUDY SCHEDULE OF EVENTS AND PROCEDURES

#### 8.1. Schedule of Events

Study assessments and procedures are presented by study period and visit in Table 1.

**Table 1:** Schedule of Events

| | Screenii<br>random | | Treatment Period | | | | | | | Fol | EOS | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Screen | Pre-<br>rand | Baseline | Wk 1 | Wk 2 | Wk 4 | Wk 8 | Wk 12 | EOT<br>Wk 16 | ET¹/<br>JR<br>Pre-<br>Op | Wk 26 | Wk 36 | ET¹ /JR Pre- Op | Wk 64 |
| Study Day | Up to 30<br>Days | 7 to 10<br>Days | 1 | 8 | 15 | 29 | 57 | 85 | 113 | | 183 | 253 | | 449 |
| Visit Window (days) | | | | ±1 | ±3 | ±7 | ±7 | ±7 | ±7 | | ±7 | ±7 | | ±7 |
| Visit/Phone Contact<br>Number | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | | Visit 10 | Visit 11 | | Phone<br>1 |
| Screening/Baseline: | | | | | | | | | | | | | | |
| Inclusion/Exclusion <sup>2</sup> | X | X | X | | | | | | | | | | | |
| Main study informed consent | X | | | | | | | | | | | | | |
| Genomics sub-study informed consent <sup>3</sup> | X | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | |
| Medication history | X | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | |
| Diary instructions | | X | X | | | | | | | | | | | |
| Training on pain reporting /patient education brochures <sup>4</sup> | X | X | | | | | | | | | | | | |
| MRI for index joint,<br>contralateral joint & any<br>hip or knee with K-L ≥3 | X | | | | | | | | | | | | | |
| Randomization | | | X | | | | | | | | | | | |
| Treatment: | | | | | | | | | | | | | | |
| Discontinue non-study pain medications | | X | | | | | | | | | | | | |
| Study drug SC injection <sup>5</sup> | | | X | | | X | X | X | | | | | | |
| Dispense to home paracetamol/acetaminophen | | X | X | | | X | X | X | | | | | | |
| Paracetamol/<br>acetaminophen<br>accountability | | | X | | X | X | X | X | X | X | | | | |
| Record rescue medication use in diary <sup>6</sup> | | X | X | X | X | X | X | X | X | X | | | | |
| Concomitant therapies | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Patient-Completed Assess | sments/Effic | acy: | | | | | | | | | | | | |
| WOMAC <sup>7, 22</sup> | X <sup>7</sup> | | X | | X | X | X | X | X | X | X | X | X | |

Regeneron Pharmaceuticals, Inc.


| | Screenii<br>random | | Treatment Period | | | | | | Fol | EOS | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Screen | Pre-<br>rand | Baseline | Wk 1 | Wk 2 | Wk 4 | Wk 8 | Wk 12 | EOT<br>Wk 16 | ET¹/<br>JR<br>Pre-<br>Op | Wk 26 | Wk 36 | ET¹ /JR - Pre- Op | Wk 64 |
| Study Day | Up to 30<br>Days | 7 to 10<br>Days | 1 | 8 | 15 | 29 | 57 | 85 | 113 | | 183 | 253 | | 449 |
| Visit Window (days) | | | | ±1 | ±3 | ±7 | ±7 | ±7 | ±7 | | ±7 | ±7 | | ±7 |
| Visit/Phone Contact<br>Number | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | | Visit 10 | Visit 11 | | Phone<br>1 |
| Neurological<br>Assessments: | | | | | | | | | | | | | | |
| Nerve conduction | $X^8$ | | | | | | X | | X | $X^9$ | | X | $X^9$ | |
| Neurological examination (full) | X | | X | | X | X | X | X | X | X | X | X | X | |
| Survey of autonomic symptoms <sup>22</sup> | X | | X | | X | X | X | X | X | X | X | X | X | |
| Orthostatic blood<br>pressure assessment and<br>heart rate <sup>10,11</sup> | X | X | X | | X | X | X | X | X | X | X | X | X | |
| Safety: | | | | | | | | • | | | • | • | | |
| Vital signs <sup>11</sup> | X | | X | | X | X | X | X | X | X | X | X | X | |
| Electrocardiogram | X | | | | | | | | X | X | | | | |
| Physical examination and weight | X | | | | | | | | X | X | | X | X | |
| Joint pain questionnaire <sup>22</sup> | X | | X | | X | X | X | X | X | X | X | X | X | |
| Event-triggered imaging <sup>12</sup> | | | | X | X | X | X | X | X | X | X | X | X | |
| Adverse Events | | | | | | | | | | | | | > | |
| SC injection site evaluation | | | X | | | X | X | X | | | | | | |
| Bilateral X-rays (knee, hip, shoulder) | X <sup>13</sup> | | | | | | | | X | X | | X | X | |
| Pre-op questionnaire (JR follow-up) <sup>14</sup> | | | | | | | | | | X | | | X | |
| MRI affected joint(s) -<br>AA patients only <sup>15</sup> | | | | | | | | | | | | | | X |
| End of study phone contact <sup>16</sup> | | | | | | | | | | | | | | X |
| Laboratory Testing: | | | | | | | | | | | | | | |
| Urine drug test <sup>17</sup> | X | | | | | | | | | | | | | |
| Hematology <sup>17</sup> | X | | | | | X | | X | X | X | X | X | X | |
| Blood chemistry <sup>17</sup> | X | | | | | X | | X | X | X | X | X | X | |

Regeneron Pharmaceuticals, Inc.


| | Screenii<br>random | | Treatment Period | | | | | | | Fol | EOS | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | Screen | Pre-<br>rand | Baseline | Wk 1 | Wk 2 | Wk 4 | Wk 8 | Wk 12 | EOT<br>Wk 16 | ET <sup>1</sup> / | Wk 26 | Wk 36 | ET¹ /JR Pre- Op | Wk 64 |
| Study Day | Up to 30<br>Days | 7 to 10<br>Days | 1 | 8 | 15 | 29 | 57 | 85 | 113 | JR | 183 | 253 | | 449 |
| Visit Window (days) | | | | ±1 | ±3 | ±7 | ±7 | ±7 | ±7 | Pre-<br>Op | ±7 | ±7 | | ±7 |
| Visit/Phone Contact<br>Number | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | | Visit 10 | Visit 11 | | Phone 1 |
| Urinalysis and urine electrolytes <sup>17</sup> | X | | | | | X | | X | X | X | X | X | X | |
| ESR | X | | | | | | | | | | | | | |
| HbA1c <sup>17</sup> | X | | | | | | | | | | | | | |
| FSH and estradiol <sup>17,18</sup> | X | | | | | | | | | | | | | |
| Pregnancy test (for WOCBP) <sup>19</sup> | X -<br>Serum | | X -<br>Urine | | | X -<br>Urine | X -<br>Urine | X -<br>Urine | X -<br>Urine | X –<br>Urine | X -<br>Urine | X –<br>Urine | X –<br>Urine | |
| PK, Antibody, and Resea | rch Samples | s <b>:</b> | | | | | | | | | | | | |
| PK sample <sup>20</sup> | | | X | X | X | X | X | X | X | X | | X | X | |
| ADA samples <sup>20</sup> | | | X | | | | | | X | X | | X | X | |
| Genomics sub-study sample (optional) <sup>3</sup> | | | X | | | | | | | | | | | |
| hs-CRP sample <sup>20,21</sup> | | | X | | | X | | | X | X | | X | X | |
| Research serum/plasma sample <sup>20,21</sup> | | | X | | | X | | | X | X | | X | X | |

AA: Adjudicated arthropathy ADA: Anti-drug antibody EOS: End of study EOT: End of treatment

ESR: Erythrocyte sedimentation rate

ET: Early termination

FSH: Follicle stimulating hormone HbA1c: Glycated hemoglobin

hs-CRP: high-sensitivity C-reactive Protein

JR: Joint replacement

MRI: Magnetic resonance imaging

PK: Pharmacokinetic Pre-op: Pre-operative Pre-rand: Pre-randomization

SC: Subcutaneous Wk: Week

WOCBP: Women of childbearing potential

WOMAC: Western Ontario and McMaster Universities Osteoarthritis Index

#### 8.1.1. Footnotes for the Schedule of Events Table 1

- 1. Patients who discontinue study drug will be encouraged to follow the visit schedule throughout the entire study. If a patient chooses to end study participation he/she will be asked to return to the study site as soon as possible for an early termination visit. Imaging assessments need to be repeated if it has been >30 days since the joints were last imaged. If it has been ≤30 days since imaging assessments were completed, imaging assessments may be completed at the discretion of the investigator.
- 2. HIV and/or hepatitis testing will be performed on a country-by-country basis, according to local guidelines if required by regulatory authorities or ethics boards. Patients must complete all other inclusion/exclusion assessments before undergoing the nerve conduction assessments.
- 3. Only for patients who provide written informed consent for the optional genomics sub-study. The sample should be collected at the day 1 (baseline/randomization) visit, but may be collected at any visit during the study after a patient has been randomized.
- 4. At the screening and pre-randomization visits, study staff will review the "Participating in a Research Study: What You Need to Know" brochure and the "Reporting Your Pain" brochure with patients to ensure they understand what a clinical study is and how to report their pain accurately. At subsequent visits, patients will be asked to review the 'Reporting Your Pain' brochure themselves. At any time during the conduct of the study, patients may require retraining by study staff.
- 5. Study drug administration will be the last procedure at each dosing visit, and will be administered after all laboratory, PK, ADA, and research samples have been collected and all study related activities have been performed. Patients will be observed in the clinic for approximately 1 hour after SC study drug is administered.
- 6. Use of study-provided rescue medication will be recorded daily using diaries. Acetaminophen/paracetamol use will be reported from pre-randomization visit to week 16.
- 7. The WOMAC pain sub-scale will be evaluated for both knees and both hip joints at the screening visit only. Then, the WOMAC Full Survey will be completed only for the index joint at the subsequent visits.
- 8. Nerve conduction can be performed during screening or pre-randomization. Patients must complete all other inclusion/exclusion assessments before undergoing the nerve conduction assessments. Randomization cannot occur until there is confirmation from the central reader assessment that the results are within the established parameters.
- 9. Nerve conduction assessments should be performed at the early termination visit if it has been >2 weeks since the last nerve conduction assessment.
- 10. Blood pressure measurements to assess for orthostatic hypotension may be discontinued following regulatory approval if the safety database does not reveal an imbalance for the fasinumab-treated patients.

- 11. If the pulse is less than 45 bpm at any visit, an ECG with rhythm strip will be obtained and sent to the central reader to confirm the heart rate and rhythm.
- 12. Imaging (X-ray and/or MRI) will be performed at the investigator's discretion on any joint with worsening or exacerbation of pain beyond the fluctuations in pain typical for that patient's OA. This imaging will be submitted to the adjudication committee for review.
- 13. If screening radiographs are inconclusive for potential joint related findings, an MRI must be performed. Confirmation from the central reader that there are no exclusionary findings on the MRI must be received before a patient can be randomized.
- 14. In the event that a patient must undergo JR surgery during the study, the patient must complete the pre-operative visit (early termination assessments, as applicable) and the procedures outlined in the schedule of events for JR follow-up. This will include a Knee Society Score questionnaire for knee replacements or Harris Hip Score questionnaire for hip replacements. The pre-operative visit must be completed before the JR surgery. Pre-operative images will be submitted to the adjudication committee for review.
- 15. If the AA joint(s) has undergone JR, an X-ray may be substituted for an MRI.
- 16. The purpose of this phone contact is to ask the patient if he/she has had or is scheduled (or on a waiting list) to have JR surgery. Pre-operative images will be submitted to the central reader for adjudication, if available.
- 17. Samples will be analyzed by the central laboratory and results will be evaluated by the investigator.
- 18. Assessment of follicle-stimulating hormone (FSH) and estradiol levels are only to be performed if assessment of postmenopausal status is required (ie, for female patients ≤59 years of age).
- 19. In the event of a positive urine pregnancy test result, the patient must have a serum pregnancy test with a negative result in order to continue study drug. If the serum pregnancy test is positive, the patient must be withdrawn from study drug and should be asked to return to the clinic for all remaining study visits per the visit schedule.
- 20. Collection of samples for PK, ADA, and research are mandatory at the time points specified above. In addition, PK, ADA, and research samples may be drawn at any scheduled visit or unscheduled visit if a patient experiences a treatment-related safety TEAE. Samples should be collected prior to study drug administration on study drug dosing days.
- 21. Biomarker samples should be collected after the patients have been fasting overnight or for 8 hours (in the event of an afternoon visit).
- 22. Patient-reported outcome measures should be completed before any clinical assessments.

Table 2: Follow-up Period for Patients Undergoing Joint Replacement Surgery on Study

| | Post-Operative Follow-up Visit 1 4 weeks after joint replacement surgery | Long-Term Follow-up Visit 2 20 weeks after joint replacement surgery |
|---|---|---|
| Follow-up Study Day (Visit Window) <sup>1</sup> | Follow-up Day 29 (±5) | Follow-up Day 140 (±7) |
| Treatment: | | |
| Concomitant medications and therapy | X | X |
| Safety: | | |
| Adverse events | | → |
| Vital signs | X | X |
| Orthostatic blood pressure <sup>2</sup> | X | X |
| Physical examination with joint examination | X | X |
| Medical history related to the joint replacement | X | X |
| Joint pain questionnaire | X | X |
| Post-operative questionnaire <sup>3</sup> | X | X |
| Bilateral X-rays (shoulders, hips, knees) <sup>4</sup> | X <sup>5</sup> | X |
| Event-triggered imaging <sup>6</sup> | X | X |

## 8.1.2. Footnotes for Table 2 - Follow-up Period for Patients Undergoing Joint Replacement Surgery

- 1. All available information for patients who undergo JR surgery must be collected, including placement of the prosthesis, healing of the surgical wound and the results of the histopathologic examination.
- 2. If it is not possible to obtain orthostatic blood pressure following JR then blood pressure and pulse should be recorded.
- 3. A Knee Society Score questionnaire for knee replacements or Harris Hip Score questionnaire for hip replacements.
- 4. In the event of more than 1 JR, imaging assessments should be repeated if it has been >60 days since the joints were last imaged. If it has been ≤60 days since imaging assessments were completed, imaging assessments may be completed at the discretion of the investigator. An MRI may be requested by the imaging vendor after review of the X-rays.
- 5. Imaging will be done at week 4 if not done pre-operatively.
- 6. Imaging may be performed on any joint following a report of clinically significant worsening or exacerbation of pain in that joint.

## **8.1.3.** Early Termination Visit

Patients who are withdrawn from study drug early should be encouraged to continue in the study and complete all other study assessments without receiving study drug. If a patient decides to completely withdraw from the study, every attempt should be made to have the patient complete an early termination visit (as outlined in Table 1). Imaging assessments need to be repeated if it has been >30 days since the joints were last imaged. If it has been  $\le 30$  days since imaging assessments were completed, imaging assessments may be completed at the discretion of the investigator.

#### 8.1.4. Unscheduled Visits

All attempts should be made to keep patients on the study schedule. Unscheduled visits may be necessary to repeat testing following abnormal laboratory results, for follow-up of AEs, or for any other reason, as warranted.

## 8.2. Study Procedures

## 8.2.1. Procedures Performed Only at the Screening/Baseline Visit

The following procedures will be performed at the screening visit for the sole purpose of determining study eligibility or characterizing the baseline population:

## 8.2.1.1. Main Study Informed Consent

All patients must sign and date the Institutional Review Board (IRB)/Ethics Committee (EC)-approved written informed consent form (ICF) before study procedures are performed, per Section 14.2.

## 8.2.1.2. Genomics Sub-study Informed Consent

Patients who are willing to participate in the Genomics Sub-study, which is optional, will sign the consent form prior to the collection of samples. Samples for DNA extraction should be collected on day 1/baseline (pre-dose), but may be collected at any study visit.

#### 8.2.1.3. Medical History

The investigator or designee will take a complete medical history that includes information on concurrent medical conditions and the severity for each condition that has not resolved. This history will include a patient's history of surgical procedures.

#### **8.2.1.4.** Medication History

The investigator or designee will query patients on the medication(s) they have taken. This includes medication taken for their pain due to OA (medication history), including information on their ability to tolerate the medication, and will record the information on an electronic case report form (eCRF) for this purpose.

## 8.2.1.5. Demographics

A patient's demographic characteristics will be recorded, including age, height, weight, gender, race, and ethnicity.

#### 8.2.1.6. Determination of Osteoarthritis

Diagnosis of OA of the knee or hip will be based on the American College of Rheumatology criteria with radiologic evidence of OA (K-L score ≥2).

In addition, diagnosis of OA of the hip and knee will use the following criteria:

#### *Hip*

The American College of Rheumatology clinical and radiographic criteria for the diagnosis of OA of the hip (Altman 1991) should be used to confirm a diagnosis of OA of the hip, as applicable, at screening. The criteria consist of the following combinations:

- Hip pain, and
- At least 2 of the following 3 features:
  - Erythrocyte sedimentation rate (ESR) <20 mm/hour
  - Radiographic femoral or acetabular osteophytes
  - Radiographic joint space narrowing (superior, axial, and/or medial)

Additional information is provided in the study reference manual.

#### Knee

The American College of Rheumatology clinical and radiographic criteria for the diagnosis of OA of the knee (Altman 1986) should be used to confirm a diagnosis of OA of the knee, as applicable, at screening. The criteria consist of the following combinations:

- Knee pain
- Osteophytes on radiograph
- At least 1 of the following 3 features:
  - Age > 50 years
  - Stiffness <30 minutes</li>
  - Crepitus

Additional information is provided in the study reference manual.

## 8.2.1.7. Assessment of Childbearing Potential

Each female patient should be evaluated for childbearing potential.

Women will be considered to be of childbearing potential unless they are postmenopausal, or have had a tubal ligation, a bilateral oophorectomy, bilateral salpingectomy, or complete hysterectomy.

For women  $\ge 60$  years of age, postmenopausal is defined as at least 12 continuous months of spontaneous amenorrhea. In women  $\le 59$  years of age, postmenopausal is defined as at least

12 continuous months of spontaneous amenorrhea, with serum FSH levels >40 IU/L (>40 mIU/mL) and serum estradiol levels <5 ng/dL (<184 pmol/L) (Section 8.2.4.8).

## 8.2.1.8. Diary Training

At the screening and pre-randomization visits, patients will be trained on the use of the diary to report their daily acetaminophen/paracetamol use for OA and other non-OA-related reasons. Retraining should occur as needed throughout the conduct of the study.

#### **8.2.1.9.** Patient Education Brochures

At the screening and pre-randomization visits, study staff will review the "Participating in a Research Study: What You Need to Know" brochure and the "Reporting Your Pain" brochure with patients to ensure they understand what a clinical study is and how to report their pain accurately. At subsequent visits, patients will be asked to review the 'Reporting Your Pain' brochure themselves. At any time during the conduct of the study, patients may require retraining by study staff.

## 8.2.2. Patient-Completed Assessments and Efficacy Procedures

#### 8.2.2.1. Western Ontario and McMaster Universities Osteoarthritis Index

The WOMAC index is used to assess patients with OA of the hip or knee using 24 parameters and reported using a numerical rating scale. This index can be used to monitor the course of a disease or to determine effectiveness of study drugs. The WOMAC pain sub-scale will be evaluated for both knees and both hip joints at the screening visit. Then, patients will complete the WOMAC Full Survey on the index joint at the subsequent visits, as indicated in Table 1. If possible, the assessment should be administered and entered by the same person throughout the study.

The WOMAC index is a patient-reported outcome measure and should be completed along with other patient-reported outcome measures, but before any clinical assessments.

A copy of WOMAC assessments will be provided in the study reference manual.

#### 8.2.3. Neurological Assessments

#### 8.2.3.1. Nerve Conduction

Nerve conduction velocities and evoked amplitudes of the peroneal motor, sural sensory and ulnar sensory nerves will be assessed at the time points indicated in Table 1. Motor nerve conduction is evaluated by electrical stimulation of the nerve and recording the compound muscle action potential from surface electrodes overlying a muscle supplied by the nerve (Mallik 2005). Sensory nerve conduction is evaluated by electrically stimulating sensory fibers and recording the nerve action potential at a point further along that nerve (Mallik 2005). Data will be interpreted by a central reader. Complete guidance on how to perform the nerve conduction assessments and how to report the findings is provided in the study reference manual.

#### 8.2.3.2. Neurological Examination (Full)

A full neurological examination will be performed at the time points indicated in Table 1. Neurological findings at baseline that are not exclusionary should be recorded in the medical history. Findings at subsequent visits will be assessed by the investigator to determine if these should be recorded as an AE.

The neurological examination will cover the following domains: motor, sensory, cranial nerves, reflexes, and coordination/balance and assessment for presence/absence of signs of carpal tunnel syndrome and may be conducted by any clinician at the site qualified to do so. Whenever possible, the same clinician who conducts the baseline neurological examination should continue to conduct the examinations on a given patient. The investigator may refer patients with persistent or worsening neurologic symptoms for a neurologic consultation, if clinically indicated. Additional neurologic assessments may include other tests as deemed clinically necessary in the judgement of the neurologist.

Complete guidance on how to conduct the full neurologic examination is provided in the study reference manual.

## 8.2.3.3. Survey of Autonomic Symptoms

The survey of autonomic symptoms will be completed by the patient at the time points indicated in Table 1. The completed survey will be reviewed for signs and symptoms of autonomic dysfunction by the investigator/medical designee at each visit prior to study drug injection at the time points indicated in Table 1. If possible, the assessment should be completed by the same person throughout the study. A patient report of having experienced symptoms of autonomic dysfunction will serve as a tool to prompt further evaluations as deemed necessary by the investigator or medical designee.

Survey of Autonomic Symptoms is a patient-reported outcome measure and should be completed along with other patient-reported outcome measures, but before any clinical assessments.

A copy of the survey is provided in the study reference manual.

#### 8.2.3.4. Orthostatic Blood Pressure Assessment and Heart Rate

An assessment of orthostatic blood pressure will be conducted at the time points indicated in Table 1. The assessments should be conducted as per the instructions in the study manual. A patient will be determined to have orthostatic hypotension if any of the following criteria are met:

If the supine systolic blood pressure is <160 mm Hg, a decrease in either the 1 or 3 minute standing systolic blood pressure of  $\ge 20$  mm Hg or a decrease in the standing diastolic blood pressure of  $\ge 10$  mm Hg from the supine systolic or diastolic blood pressure, respectively

OR

If the supine systolic blood pressure is  $\geq 160$  mm Hg, a decrease in either the 1 or 3 minute standing systolic blood pressure of  $\geq 30$  mm Hg or a decrease in the standing diastolic blood pressure of  $\geq 15$  mm Hg from the supine systolic or diastolic blood pressure, respectively

OR

An increase in either the 1 or 3 minute standing heart rate of ≥30 bpm from the supine heart rate

OR

The patient is unable to stand for either one of the standing blood pressure measurements due to dizziness or lightheadedness

If the initial assessment for orthostatic hypotension is consistent with the above definition, the supine and standing blood pressures and/or pulse should be repeated as outlined above, up to 2 more times.

Refer to Section 9.6.1.2 for details on referral to specialists and reporting.

#### 8.2.4. Safety Procedures

## **8.2.4.1.** Vital Signs

Vital signs, including body temperature and respiratory rate, will be collected pre-dose at time points according to Table 1. Blood pressure and heart rate will be collected as part of the orthostatic hypotension assessments. If at any visit after the randomization visit the pulse is less than 45 bpm, an ECG with rhythm strip will be obtained to confirm the heart rate and rhythm.

## 8.2.4.2. Electrocardiogram

A standard 12-lead ECG will be performed at the time points indicated in Table 1, with the patient in the supine position for approximately 5 minutes and prior to blood samples being drawn. Heart rate will be recorded from the ventricular rate, and the PR, QRS, and the QT and QTc intervals will be recorded. The ECG data will be read by a central reading center. Detailed procedures will be provided in a separate manual provided by the central reading center.

## 8.2.4.3. Physical Examination and Body Weight

A thorough and complete physical examination will be performed at time points according to Table 1. Body weight will also be measured. Care should be taken to examine and assess any abnormalities that may be present, as indicated by the patient's medical history.

## 8.2.4.4. Joint Pain Questionnaire

A joint pain questionnaire will be completed by the patient at the time points indicated in Table 1. For each knee, hip, and shoulder joint, the patient will be prompted to indicate if he or she has experienced pain. A patient report of having experienced pain will serve as a tool to prompt further evaluations as deemed necessary by the investigator.

Joint Pain Questionnaire is a patient-reported outcome measure and should be completed along with other patient-reported outcome measures, but before any clinical assessments.

A copy of the assessment is provided in the study reference manual.

## **8.2.4.5. Imaging**

Radiographs of the large joints (knees, hips, and shoulders) will be taken using a standard approach at the time points indicated in Table 1. An MRI of the index and contralateral joints must be performed at screening. Magnetic resonance imaging will also be performed on any hip or knee joint with a K-L score of  $\geq 3$ . Radiographs and an MRI must be performed on any joint following

a report of clinically significant worsening or exacerbation of pain in that joint. An X-ray and an MRI should also be performed pre-operatively if a patient is to have a JR during the study. Event based and pre-operative images will be submitted for adjudication. Detailed procedures will be provided in a separate manual provided by the central imaging center. Radiograph or MRI will be sent to a central reader, where the images will be digitized.

#### Radiographs

Weight-bearing (standing) posterior-anterior radiographs of both knees in the semi-flexed position, and anterior-posterior radiographs of both hips and both shoulders, will be conducted at these visits. Additional instructions for positioning of joints are provided in the study reference manual.

Radiographs of the knees, hips, and shoulders will be sent to a central reader and evaluated to confirm no evidence of AA such as rapidly progressive osteoarthritis type 1 or 2, subchondral insufficiency fracture, or osteonecrosis.

## **MRI**

During screening, MRIs of the index and contralateral joints as well as joints with a K-L score ≥3 will be sent to a central reader to confirm that there is no evidence of exclusionary features. Confirmation that there are no exclusionary findings on MRI must be received before a patient can be randomized. An MRI of any joint will be considered if radiographs taken after randomization suggest the presence of an abnormal process inconsistent with normal progression of OA, as determined by the investigator or central reader.

At the end of study phone contact, patients who had an AA will have an MRI performed of the affected joint(s). If the affect joint has undergone JR, an X-ray may be substituted for an MRI.

Refer to the supplemental imaging manuals for data collection and management procedures.

#### 8.2.4.6. End of Study Phone Contact and Additional Imaging

An end of study phone contact will be conducted at 52 weeks following the last dose of study drug. Patients will be asked whether they underwent JR surgery following the last in-clinic visit of the follow-up period or whether they are scheduled (or on a waiting list) for JR surgery. Patients who had JR surgery will also be asked to submit pre-operative imaging (X-ray and MRI, if available) for adjudication. Patients who had an AA will have an MRI performed of the affected joint(s). If the affected joint has undergone JR, an X-ray may be substituted for an MRI.

## 8.2.4.7. Procedures to be Performed Only in the Event of a Joint Replacement Surgery

In the event that a patient must undergo JR surgery during the treatment or follow-up periods, the patient will be discontinued from study drug and asked to return for a pre-operative visit. The pre-operative visit should be completed before JR surgery if possible, and pre-operative images will be submitted to the adjudication committee for review. Following the JR surgery, the patient will complete follow-up safety evaluations at 4 weeks and 20 weeks after surgery (see Table 2).

In the event that the pre-operative visit is not performed, standard-of-care pre-operative images of the joint with JR must be obtained and submitted to the central imaging vendor's adjudication committee for review. Imaging of all other joints per the pre-operative visit procedures will be done post-operatively at the first JR follow-up study visit (4 weeks after surgery) if not done before surgery.

All available medical history/information for patients who undergo JR surgery must be collected, including the results of histopathologic examination.

Full details of these assessments are provided in the study reference manual.

## **Knee Society Score**

The Knee Society Score is an investigator-completed questionnaire that is used to objectively measure a patient's ability to function before and after total knee arthroplasty (Insall 1989). If possible, the assessment should be completed by the same person throughout the study.

## Harris Hip Score

The Harris Hip Score is an investigator-completed questionnaire that is used to objectively measure a patient's ability to function before and after total hip arthroplasty (Harris 1969). If possible, the assessment should be completed by the same person throughout the study.

## 8.2.4.8. Laboratory Testing

The central laboratory will analyze all screening and on-study laboratory samples for blood chemistry, hematology, HbA1c, urine analysis, urine drug tests, and serum pregnancy tests. Urine pregnancy and ESR testing will be done at the site using kits provided by the central laboratory.

Regeneron or its designee will be responsible for fasinumab PK, anti-fasinumab antibody, biomarker development, and pharmacogenetic sample assessments; the central laboratory will ship the samples to Regeneron or a specialty laboratory depending on the assessment.

All samples will be collected before study drug administration. Missed tests should be reported in the source documents and in the eCRF, as appropriate. Central laboratory kits will be provided for sample collection and shipment. Detailed instructions for blood sample collection are in the laboratory manual provided to study sites.

Samples for laboratory testing will be collected at time points according to Table 1. Tests will include:

#### **Blood Chemistry**

SodiumTotal protein, serumTotal bilirubinPotassiumCreatininePhosphorusChlorideBlood urea nitrogenUric acid

Carbon dioxide Aspartate aminotransferase (AST) Creatine phosphokinase

Calcium Alanine aminotransferase (ALT)

Glucose Alkaline phosphatase
Albumin Lactate dehydrogenase

#### Hematology

Hemoglobin Differential:
Hematocrit Neutrophils
Red blood cells (RBCs) Lymphocytes
White blood cells (WBCs) Monocytes
Red cell indices Basophils
Platelet count Eosinophils

#### Urinalysis

Color Glucose RBC

Clarity Blood Hyaline and other casts

pH Bilirubin Bacteria
Specific gravity Leukocyte esterase Epithelial cells
Ketones Nitrite Crystals
Protein WBC Yeast

#### Urine Electrolytes

Creatinine Phosphorus

#### Other Laboratory Tests

Serum and urine samples for pregnancy testing will be collected from women of childbearing potential (WOCBP) (as defined in Section 8.2.1.7) at time points according to Table 1. At dosing study visits, urine pregnancy testing will be done before the study drug is administered. In the event of a positive urine pregnancy test result, the patient should have a serum pregnancy test with a negative result in order to continue study drug. If the serum pregnancy test is positive, the patient should be withdrawn from study drug and should be asked to return to the clinic for all remaining study visits per the visit schedule (see Table 1).

To assess postmenopausal status for women ≤59 years of age, serum samples to test for FSH levels and estradiol levels will be collected for analysis at the central laboratory according to Section 8.2.1.7.

Samples will be collected for HbA1c and ESR testing at time points according to Table 1.

Urine drug testing will be performed at screening and includes amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates.

Blood samples for study drug PK and ADA assessment (Section 8.2.5) will also be collected.

## Abnormal Laboratory Values and Laboratory Adverse Events

All laboratory values must be reviewed by the investigator or authorized designee.

Significantly abnormal test results that occur after start of treatment must be repeated to confirm the nature and degree of the abnormality. When necessary, appropriate ancillary investigations should be initiated. If the abnormality fails to resolve or cannot be explained by events or conditions unrelated to the study medication or its administration, the medical monitor must be consulted.

The clinical significance of an abnormal test value, within the context of the disease under study, must be determined by the investigator.

Criteria for reporting laboratory values as an AE are provided in Section 9.4.5. Evaluation of severity of laboratory abnormalities will be assessed according to the scale outlined in Section 9.5.1.

## **8.2.4.9.** Injection Site Evaluations

An injection site evaluation should be conducted following the injection at each dosing visit, according to Table 1.

## 8.2.5. Pharmacokinetic and Anti-Drug Antibody Procedures

#### 8.2.5.1. Drug Concentration Measurements and Samples

Samples for drug concentration will be collected at time points listed in Table 1. Detailed instructions for blood sample collection are included in the laboratory manual provided to study sites.

Any unused samples may be used for exploratory biomarker research.

## 8.2.5.2. Anti-Drug Antibody Measurements and Samples

Samples for ADA assessment will be collected at time points listed in Table 1. Detailed instructions for blood sample collection are included in the laboratory manual provided to study sites.

Any unused samples may be used for exploratory biomarker research.

#### 8.2.6. Research Samples

#### 8.2.6.1. Biomarkers

Serum and plasma samples will be collected at time points according to Table 1. These samples may be used to measure biomarkers related to inflammation, collagen and bone turnover, OA pain and NGF and may include CTX-I, osteocalcin, high-sensitivity C-reactive protein and matrix

metalloprotein generated collagen fragments (CIM, C3M). Samples may be used to study other markers of collagen and bone turnover, OA and pain. If necessary, samples may also be used to identify markers associated with AEs.

#### **8.2.6.2.** Future Biomedical Research

Unused research samples, as well as unused PK and ADA samples, will be stored for up to 15 years after the final date of the database lock. The unused samples may be utilized for future biomedical research of OA and other diseases. No additional samples will be collected for future biomedical research. After 15 years, any remaining samples will be destroyed.

## 8.2.6.3. Genomics Sub-study - Optional

Patients who agree to participate in the genomics sub-study will be required to sign a separate genomics sub-study ICF before collection of the samples. Patients are not required to participate in the genomics sub-study in order to enroll in the primary study. Samples for DNA extraction should be collected on day 1/baseline (pre-dose), but may be collected at any study visit.

DNA samples for the genomics sub-study will be double-coded as defined by the International Council for Harmonisation (ICH) guideline E15. Sub-study samples will be stored for up to 15 years after the final date of the database lock and may be used for research purposes. The purpose of the genomic analyses is to identify genomic associations with collagen and bone turnover, OA, pain, and response to fasinumab. In addition, associations between genomic variants and prognosis or progression of OA as well as other diseases may also be studied. These data may be used or combined with data collected from other studies to identify and validate genomic markers related to the study drug or other diseases. Analyses may include sequence determination or single nucleotide polymorphism studies of candidate genes and surrounding genomic regions. Other methods, including whole-exome sequencing, whole-genome sequencing, and DNA copy number variation may also be performed. The list of methods may be expanded to include novel methodology that may be developed during the course of this study or sample storage period.

The results of these future biomedical research analyses will not be presented in the clinical study report.

## 9. SAFETY DEFINITIONS, REPORTING, AND MONITORING

# 9.1. Obligations of Investigator

The investigator must promptly report to the IRB or EC all unanticipated problems involving risks to patients, according to local regulations. This may include death from any cause and all serious adverse events (SAEs) related to the use of the study drug. It is recommended that all SAEs be reported to the IRB or EC according to local regulations.

## 9.2. Obligations of Sponsor

During the course of the study, the sponsor will report in an expedited manner all SAEs that are both unexpected and at least reasonably related to the study drug (SUSAR), to the health authorities, EC/IRBs as appropriate, and to the investigators (in a blinded manner).

Any AE not listed as an expected event in the Reference Safety Information section of the Investigator's Brochure will be considered unexpected. Any worsening of or new onset of symptoms related to OA that occur during the screening period prior to study drug administration will be considered expected.

In addition, the sponsor will report all other SAEs to the health authorities, according to local regulations.

At the completion of the study, the sponsor will report all safety observations made during the conduct of the trial in the clinical study report to health authorities and ECs/IRBs as appropriate.

## 9.3. **Definitions**

#### 9.3.1. Adverse Event

An AE is any untoward medical occurrence in a patient administered a study drug which may or may not have a causal relationship with the study drug. Therefore, an AE is any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease which is temporally associated with the use of a study drug, whether or not considered related to the study drug.

An AE also includes any worsening (ie, any clinically significant change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the study drug.

#### 9.3.2. Serious Adverse Event

An SAE is any untoward medical occurrence that at any dose:

- Results in **death** includes all deaths, even those that appear to be completely unrelated to study drug (eg, a car accident in which a patient is a passenger).
- Is **life-threatening** in the view of the investigator, the patient is at immediate risk of death at the time of the event. This does not include an AE that had it occurred in a more severe form, might have caused death.
- Requires in-patient hospitalization or prolongation of existing hospitalization. In-patient hospitalization is defined as admission to a hospital or an emergency room for longer than 24 hours. Prolongation of existing hospitalization is defined as a

hospital stay that is longer than was originally anticipated for the event, or is prolonged due to the development of a new AE as determined by the investigator or treating physician.

- Results in persistent or significant **disability/incapacity** (substantial disruption of one's ability to conduct normal life functions).
- Is a congenital anomaly/birth defect
- Is an **important medical event** Important medical events may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the patient or may require intervention to prevent one of the other serious outcomes listed above. Examples of these include intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

Criteria for reporting SAEs must be followed for these events. See Section 9.4 for more information on recording and reporting SAEs.

## 9.3.3. Adverse Events of Special Interest

An AESI (serious or non-serious) is one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate. Such an event might warrant further investigation in order to characterize and understand it. Depending on the nature of the event, rapid communication by the trial sponsor to other parties (eg, regulators) might also be warranted (Section 9.4.3).

# 9.4. Recording and Reporting Adverse Events

#### 9.4.1. Adverse Events

The investigator (or designee) will record all AEs that occur from the time the informed consent is signed until the end of the follow-up period (week 36)/early termination visit. Refer to the study reference manual for the procedures to be followed.

Information on follow-up for AEs is provided in Section 9.4.6. Laboratory, vital signs, or ECG abnormalities are to be recorded as AEs as outlined in Section 9.4.5.

#### 9.4.2. Serious Adverse Events

All SAEs, regardless of assessment of causal relationship to study drug, must be reported to the sponsor (or designee) within 24 hours. Refer to the study reference manual for the procedure to be followed.

Information not available at the time of the initial report must be documented in a follow-up report. Substantiating data such as relevant hospital or medical records and diagnostic test reports may also be requested.

In the event the investigator is informed of an SAE after the patient completes the follow-up period (week 36)/early termination visit, the following will apply:

- SAE with an onset within 30 days of the end of the follow-up (week 36)/early termination visit the SAE will be reported to the sponsor. The investigator should make every effort to obtain follow-up information on the outcome until the event is considered chronic and/or stable.
- SAE with an onset day greater than 30 days from the end of follow-up period (week 36)/early termination visit only SAEs deemed by the investigator to be drug-related will be reported to the sponsor. The investigator should make every effort to obtain follow-up information on the outcome of a drug-related SAE until the event is considered chronic and/or stable.
- SAE reported by the patient at the end of the study phone call and deemed by the investigator to be drug-related will be reported to the sponsor. The investigator should make every effort to obtain follow-up information on the outcome of a drug-related SAE until the event is considered chronic and/or stable.

## 9.4.3. Other Events that Require Accelerated Reporting to Sponsor

The following events also require reporting to the sponsor (or designee) within 24 hours of learning of the event:

**Symptomatic Overdose of Study Drug:** Accidental or intentional overdose of at least 2 times the intended dose of study drug within the intended therapeutic window, if associated with an AE

**Pregnancy:** Although pregnancy is not considered an AE, it is the responsibility of the investigator to report to the sponsor (or designee), within 24 hours of identification, any pregnancy occurring in a female study patient during the study or within 20 weeks of the last dose of study drug. Any complication of pregnancy affecting a female study patient and/or fetus and/or newborn that meets the SAE criteria must be reported as an SAE. Outcome for all pregnancies should be reported to the sponsor.

Adverse Events of Special Interest: All AESI, serious and non-serious, must be reported within 24 hours of identification using the same reporting process as for SAE reporting per Section 9.4.2. Monitoring of AESIs is described in Section 9.6.1. Adverse events of special interest for this study include the following:

- Adjudicated arthropathy (as confirmed by adjudication)
- Joint replacement surgery (refer to Section 9.6.1.4 for when to report as an AESI)
- Sympathetic nervous system dysfunction (as diagnosed after consultation with an appropriate specialist, such as a neurologist and/or cardiologist)
- Peripheral sensory AEs that require a neurology or other specialty consultation

Refer to the study manual for the procedures to be followed.

## 9.4.4. Reporting Adverse Events Leading to Withdrawal from the Study

All AEs that lead to a patient's withdrawal from the study must be reported to the sponsor's Medical/Study Director within 30 days.

Refer to the study reference manual for the procedures to be followed.

## 9.4.5. Abnormal Laboratory, Vital Signs, or Electrocardiogram Results

The criteria for determining whether an abnormal objective test finding should be reported as an AE include:

- the test result is associated with accompanying symptoms, and/or
- the test result requires additional diagnostic testing or medical/surgical intervention, and/or
- the test result leads to a change in dosing (outside of protocol-stipulated dose adjustments), discontinuation from the study, significant additional concomitant drug treatment, or other therapy

Contact the Medical/Study Director in the event the investigator feels that an abnormal test finding should be reported as an AE, although it does not meet any of the above criteria.

Repeating an abnormal test, in the absence of any of the above conditions, does not constitute an AE. Any abnormal test result that is determined to be an error does not require reporting as an AE.

Evaluation of severity of laboratory abnormalities will be assessed according to the scale outlined in Section 9.5.1.

## **9.4.6.** Follow-up

Adverse event information will be collected until the patient's last study visit.

Serious adverse event information will be collected until the event is considered chronic and/or stable.

# 9.5. Evaluation of Severity and Causality

#### 9.5.1. Evaluation of Severity

The severity of AEs will be graded according to the following scale:

- **Mild:** Does not interfere in a significant manner with the patient normal functioning level. It may be an annoyance. Prescription drugs are not ordinarily needed for relief of symptoms, but may be given because of personality of the patient.
- **Moderate:** Produces some impairment of functioning but is not hazardous to health. It is uncomfortable or an embarrassment. Treatment for symptom may be needed.
- **Severe:** Produces significant impairment of functioning or incapacitation and is a definite hazard to the subject's health. Treatment for symptom may be given and/or patient hospitalized.

If a laboratory value is considered an AE, its severity should be based on the degree of physiological impairment the value indicates.

## **Injection Site Reactions**

The severity of injection site reactions will be graded according to the following scale (semi-colon indicates "or" within description of grade):

- Mild: Pain that does not interfere with activity; mild discomfort to touch; <5 cm of erythema or induration that does not interfere with activity.
- **Moderate**: Pain that requires repeated use of non-narcotic pain reliever >24 hours or interferes with activity; discomfort with movement; 5.1 cm to 10 cm erythema or induration or induration that interferes with activity.
- Severe: Pain that requires any use of narcotic pain reliever or that prevents daily activity; significant discomfort at rest; >10 cm erythema or induration; prevents daily activity; requires emergency room visit or hospitalization; necrosis or exfoliative dermatitis.

## 9.5.2. Evaluation of Causality

## Relationship of Adverse Events to Study Drug:

The relationship of AEs to study drug will be assessed by the "blinded" investigator, and will be a clinical decision based on all available information. The following question will be addressed:

Is there a reasonable possibility that the AE may have been caused by the study drug?

The possible answers are:

**Not Related:** There is no reasonable possibility that the event may have been caused by the study drug.

**Related:** There is a reasonable possibility that the event may have been caused by the study drug.

The investigator should justify the causality assessment of each SAE.

A list of factors to consider when assessing the relationship of AEs to study drug is provided below. Please note that this list is not exhaustive.

Is there a reasonable possibility that the event may have been caused by the study drug?

No:

- due to external causes such as environmental factors or other treatment(s) being administered
- due to the patient's disease state or clinical condition
- do not follow a reasonable temporal sequence following the time of administration of the dose of study drug
- do not reappear or worsen when dosing with study drug is resumed

Yes:

• could not be explained by environmental factors or other treatment(s) being administered

- could not be explained by the patient's disease state or clinical condition
- follow a reasonable temporal sequence following the time of administration of the dose of study drug
- resolve or improve after discontinuation of study drug
- reappear or worsen when dosing with study drug
- are known or suspected to be a response to the study drug based upon preclinical data or prior clinical data

## Relationship of Adverse Events to Study Conduct

The relationship of AEs to study conduct will be assessed by the "blinded" investigator, and will be a clinical decision based on all available information. The following question will be addressed:

Is there a reasonable possibility that the AE may have been caused by study conduct?

The possible answers are:

**Not Related:** There is no reasonable possibility that the event may have been caused by study conduct.

**Related:** There is a reasonable possibility that the event may have been caused by study conduct.

The investigator should justify the causality assessment of each SAE.

A list of factors to consider when assessing the relationship of AEs to study conduct is provided below. Please note that the list if not exhaustive.

Is there a reasonable possibility that the event may have been caused by the study conduct?

Is there a reasonable possibility that the event may have been caused by the study conduct?

## No:

- due to external causes such as environmental factors or other treatment(s) being administered
- due to the patient's disease state or clinical condition
- do not follow a reasonable temporal sequence following the course of the study
- do not reappear or worsen when dosing with study participation is resumed

#### Yes:

- could not be explained by environmental factors or other treatment(s) being administered
- could not be explained by the patient's disease state or clinical condition
- follow a reasonable temporal sequence following the course of the study
- resolve or improve after discontinuation from study participation.
- reappear or worsen when study participation is resumed

# 9.6. Safety Monitoring

The investigator will monitor the safety of study patient at his/her site(s) as per the requirements of this protocol and consistent with current Good Clinical Practice (GCP). Any questions or concerns should be discussed with the sponsor in a timely fashion. The sponsor will monitor the safety data from across all study sites. The Medical/Study Director will have primary responsibility for the emerging safety profile of the compound, but will be supported by other departments (eg, Pharmacovigilance and Risk Management; Biostatistics and Data Management). Safety monitoring will be performed on an ongoing basis (eg, individual review of SAEs) and on a periodic cumulative aggregate basis.

## 9.6.1. Monitoring Adverse Events of Special Interest

## 9.6.1.1. Adjudicated Arthropathy

Adjudicated arthropathy is an umbrella term that encompasses the following conditions:

- Rapidly progressive OA type 1 and 2
- Subchondral insufficiency fractures
- Primary osteonecrosis

In addition, adjudicated arthropathies will be evaluated to determine if they meet destructive arthropathy criteria.

Potential events of AA will be monitored via clinical signs and symptoms of worsening joint pain during the course of the study (eg, by applying adverse experiences, the joint pain questionnaire and imaging) as well as scheduled imaging and pre-operative imaging, if a patient requires a JR during the study.

Clinically significant worsening of joint pain during the course of this study is characterized as a worsening of pain in any joint that occurs in spite of treatment with analgesics, is in the opinion of the investigator inconsistent with the normal fluctuation of pain or progression of OA, and is at least 2 weeks duration (or less than 2 weeks if deemed clinically significant at the discretion of the investigator).

If a patient reports an increase in pain as described above, study drug administration will be withheld while imaging of the affected joint, as well as any additional imaging deemed appropriate to understand the cause of the worsening pain, is performed (Section 8.2.4.5). A decision to perform imaging after patient reported of worsening of joint pain will be documented in the respective CRF page. Images, along with any other radiographic evaluation, will be submitted to the arthropathy adjudication committee for review (Section 5.3.2). The investigator may consider aspiration of synovial fluid for further analysis such as cell count and crystal analysis.

If routine imaging suggests the presence of one of the types of AA, study drug administration will be withheld. Any additional imaging deemed appropriate will be obtained. The images, along with results of any other radiographic evaluation, will be submitted to the Adjudication Committee for review (Section 5.3.2).

If the adjudication does not confirm the presence of AA, according to the adjudication criteria, study drug may be restarted.

Study drug dosing will be permanently discontinued for patients with findings that suggest AA; the patients will be referred for orthopedic consultation. If presence of AA is confirmed by the Adjudication Committee, the case must be reported as an AESI (Section 9.3.3 and Section 9.4.3).

Any patient whose study drug is discontinued due to an AA should be encouraged to return to the clinic for all remaining study visits. If JR surgery is warranted, prior to the scheduled JR, the patient should complete the pre-operative study visit and, after the JR, should complete the week 4 and week 20 post-operative study visits (Table 2). Pre-operative images, along with any other radiographic evaluation will be submitted to the arthropathy adjudication committee for review (Section 5.3.2).

Details of data collection for adjudication of events will be provided in the adjudication charter.

## 9.6.1.2. Sympathetic Nervous System Dysfunction

Sympathetic nervous system dysfunction will be monitored throughout the study through physical examination, AE reporting, assessment of orthostatic hypotension, and the Survey of Autonomic Symptoms (Section 8.2.3.3). New onset or worsening of signs and symptoms of autonomic dysfunction will be evaluated by the investigator. Sympathetic nervous system dysfunction will only be diagnosed after consultation with an appropriate specialist, such as a neurologist and/or cardiologist.

In cases in which new or worsening symptoms consistent with SNS dysfunction are moderate to severe or are clinically significant and do not resolve or return to baseline in 2 weeks (or less at the discretion of the investigator), study drug will be withheld and the patient will be referred to a specialist. If the evaluation by the appropriate specialist does not suggest SNS dysfunction, study drug may be restarted. If the specialist's evaluation does reveal SNS dysfunction then study drug will be permanently discontinued and the case reported as an AESI (Section 9.4.3).

Orthostatic hypotension may be a manifestation of SNS dysfunction. If a patient is determined to have orthostatic hypotension, study drug should be withheld and the AE should be entered in the CRF. The following procedures should be followed:

- If the patient is symptomatic and a clinical explanation for orthostatic hypotension is identified (such as a new medication or dehydration due to exercise or illness or excessive heat exposure), study drug will be withheld, and the patient should return to the study site for an unscheduled visit in 1 to 10 days for an unscheduled assessment of orthostatic hypotension.
  - If the orthostatic hypotension has resolved, study drug may be restarted.
  - If the orthostatic hypotension has not resolved, then study drug will be withheld, and the patient will be referred to a specialist (neurologist or a cardiologist) for evaluation of sympathetic nervous system dysfunction.
    - If the specialist's evaluation does not reveal new onset SNS dysfunction, including symptoms of bradycardia (lightheadedness), orthostatic hypotension (lightheadedness on standing), syncope, absence of sweating in conditions where sweating would be expected, or if the specialist's evaluation identifies an alternative cause, such as initiation of a new

medication known to cause orthostasis, then study drug may be given at the next visit.

- If the specialist's evaluation does reveal SNS dysfunction, then study drug will be permanently discontinued and the case reported as an AESI (Section 9.4.3).
- If the patient has asymptomatic orthostatic hypotension, study drug will be withheld, and the patient should return to the study site for an unscheduled visit in 1 to 10 days for an unscheduled assessment of orthostatic hypotension.
  - If the unscheduled assessment does not reveal orthostatic hypotension then study drug may be continued.
  - If the unscheduled assessment demonstrates orthostatic hypotension then study drug will continue to be withheld until the patient has been evaluated by a specialist (neurologist or a cardiologist) for evidence of SNS dysfunction.
    - If the specialist's evaluation does not reveal new SNS dysfunction including symptoms of bradycardia (lightheadedness), orthostatic hypotension (lightheadedness on standing), syncope, absence of sweating in conditions where sweating would be expected, or if the specialist's evaluation identifies an alternative cause such as initiation of a new medication known to cause orthostasis, then study drug may be restarted.
    - If the specialist's evaluation does reveal SNS dysfunction then study drug will be permanently discontinued and the case reported as an AESI (Section 9.4.3).

## 9.6.1.3. Peripheral Sensory Adverse Events

Altered peripheral sensation (eg, paraesthesia and hypoaesthesia) is an important identified risk with fasinumab (see Investigator's Brochure) and other anti-NGF compounds. Any peripheral sensory AE that, per the investigator's judgment, requires a neurology or other specialty consultation must be reported as an AESI. If any peripheral sensory event persists for 2 months, the patient must be referred for a neurology or other specialty consultation and the event must be reported as an AESI. Refer to the study manual for further details related to reporting of peripheral sensory neuropathy AEs.

If the repeated per-protocol nerve conduction test performed on the regions of the peroneal, sural, or ulnar nerves at any post-baseline visit shows a difference from baseline of >12% (based on central reader assessment), the patient will be referred for a neurology evaluation. If the neurologist's evaluation confirms the diagnosis of peripheral neuropathy, the study drug will be permanently discontinued. Refer to the study manual for further details related to reporting of results of nerve conduction tests.

#### 9.6.1.4. Joint Replacement Surgery

Any elective JR surgery planned before completion of the ICF would be part of the exclusion criteria and would not be considered an AE.

After signing of the ICF, report JR surgery as an AESI if the JR surgery is an elective event that is not associated with a new/worsening AE.

Do not report JR surgery as an AE/AESI if the JR surgery is for the treatment of a new or worsening AE. In this case, the new or worsening AE should be the reported AE/AESI term.

An end of study phone contact will be conducted approximately 52 weeks following the last dose of study drug to evaluate the number of patients who have undergone or are scheduled for JR surgery as described in Section 8.2.4.7.

## 9.7. Investigator Alert Notification

Regeneron (or designee) will inform all investigators participating in this clinical trial, as well as in any other clinical trial using the same investigational drug, of any SAE that meets the relevant requirements for expedited reporting (an AE that is serious, unexpected based on the Investigator's Brochure or this protocol, and has a reasonable suspected causal relationship to the medicinal/study drug).

#### 10. STATISTICAL PLAN

This section provides the basis for the statistical analysis plan (SAP) for the study. The SAP may be revised during the study to accommodate amendments to the clinical study protocol and to make changes to adapt to unexpected issues in study execution and data that may affect the planned analyses. The final SAP will be issued before the database is locked.

Analysis variables are listed in Section 4.

# **10.1.** Statistical Hypothesis

No formal hypothesis testing will be performed on nerve conduction measures. The treatment difference between fasinumab and placebo in the change from baseline to week 16 in nerve conduction measures will be estimated and presented descriptively along with 95% confidence intervals.

# **10.2. Justification of Sample Size**

Approximately 180 patients will be randomized in a 1:1 ratio to fasinumab 1 mg Q4W or placebo.

With this sample size, the precision of the estimated treatment difference between fasinumab and placebo at week 16 in nerve conduction velocity is no more than 1.21 m/s with a 95% confidence level, assuming a standard deviation (SD) of 3.6 m/s. This sample size provides similar precision for the estimated treatment difference in nerve conduction amplitude assuming an SD of 3.6  $\mu$ V. The assumed SDs are estimated based on the nerve conduction results from Arezzo 2008.

Assuming a 2-sided alpha level of 0.05 and a 15% dropout rate up to week 16, an enrollment of 90 patients per group will provide at least 80% power to detect an effect size of 0.46 in the WOMAC pain and physical function subscale scores (ie, absolute treatment difference of 1.1 between fasinumab and placebo with an SD of 2.4). The assumed treatment difference and SD are based on results from study R475-PN-1227.

## 10.3. Analysis Sets

## 10.3.1. Efficacy Analysis Set

The full analysis set (FAS) includes all randomized patients and is based on the treatment allocated (as randomized). Efficacy endpoints will be analyzed using the FAS.

## 10.3.2. Safety Analysis Set

The safety analysis set (SAF) includes all randomized patients who received any study drug; it is based on the treatment received (as treated). Treatment compliance/administration and all clinical safety variables will be analyzed using the SAF.

## 10.3.3. Pharmacokinetic Analysis Set

The PK analysis set includes all treated patients who received any study drug and who had at least 1 non-missing drug concentration result following the first dose of study drug.

## 10.3.4. Anti-Drug Antibody Analysis Set

The ADA analysis set includes all treated patients who had at least 1 qualified (non-missing) post-dose ADA result following the first dose of study drug.

#### 10.4. Statistical Methods

For continuous variables, descriptive statistics will include the following information: the number of patients reflected in the calculation (n), mean, median, SD, minimum, Q1, Q3, and maximum.

For categorical or ordinal data, frequencies and percentages will be displayed for each category.

#### 10.4.1. Patient Disposition

The following will be provided:

- The total number of screened patients: met the inclusion criteria regarding the target indication and signed the ICF
- The total number of randomized patients: received a randomization number
- The total number of patients in each analysis set
- The total number of patients who discontinued the study, and the reasons for discontinuation
- A listing of patients treated but not randomized, patients randomized but not treated, and patients randomized but not treated as randomized
- A listing of patients prematurely discontinued from treatment, along with reasons for discontinuation

#### **10.4.2.** Demography and Baseline Characteristics

Demographic and baseline characteristics will be summarized descriptively by treatment group, and by all patients combined.

#### 10.4.3. Efficacy Analysis

The efficacy variables will be analyzed using multiple imputation approach with mixed-effect model for repeated measure (MMRM) based on the FAS with adjustment for missing data due to lack of efficacy or AEs assuming the scores would on average return to baseline values. The imputed data for patients discontinued from study drug due to lack of efficacy or AEs will be centered at the mean baseline value. The missing data for patients discontinued from treatment due to other reasons will be imputed under missing-at-random assumption.

Missing data will be imputed 50 times to generate 50 complete data sets. Each imputed data set will be analyzed using the MMRM with terms for baseline score corresponding to the efficacy variable being analyzed, randomization strata (K-L category [2 to 3, or 4] and index joint [knee, hip]), treatment, visit, and treatment-by-visit interaction. The MMRM will be performed with an unstructured covariance matrix to model the within-patient errors. Denominator degrees of freedom will be estimated using Kenward-Roger's approximation. The results from the 50 analyses will be combined using Rubin's formulae. The least-squares mean estimates for the mean change from baseline to week 16, as well as the difference of the estimates between fasinumab and placebo with their corresponding standard errors and associated 95% confidence intervals, will be provided.

For analysis of categorical variables, eg, proportions of patients with  $\geq 30\%$  improvement in the WOMAC pain subscale scores at week 16, the Cochran Mantel Haenszel approach stratified by the randomization strata will be used with missing data considered as non-response.

## 10.4.4. Safety Analysis

Safety data including nerve conduction measures, TEAEs and treatment emergent AESIs, vital signs, physical exams, laboratory tests, ECGs, and ADA formation will be listed and summarized by treatment group.

Thresholds for potentially clinically significant values (PCSVs) in laboratory parameters and vital signs will be defined by the sponsor and be in effect at the time of final SAP approval.

The time interval to detect any AEs, including AESIs, is between the first dose of double-blinded study drug injection and the week 36 visit, as well as study drug-related SAEs occurring between the week 36 visit and the end of study.

For safety variables, 3 observation periods are defined:

- The pretreatment period is defined as the time from signing the ICF to before the first dose of study drug.
- The treatment period is defined as the day from first dose of study drug through the day of last dose (week 12) + 4 weeks.
- The follow-up period is defined from the end of on-treatment period to the week 36 visit.

## 10.4.4.1. Primary Safety Analysis

The variables for the evaluation of peripheral nerve function are the change from baseline to week 16 in the amplitude and velocity from the 3 individual nerve conduction tests.

The nerve conduction variables will be analyzed using an MMRM approach based on the safety analysis set. The model will include baseline value, randomization strata, treatment, visit, and treatment-by-visit interaction. The least-squares mean estimates for the mean change from baseline to week 16, as well as the differences of the estimates between fasinumab and placebo, with their corresponding standard errors and associated 95% confidence intervals, will be provided descriptively. Missing data due to no response or outside of test detection limit will be imputed using the first percentile of all non-missing values for that measurement prior to the MMRM analysis. Additional analysis based on observed data with no imputation may also be performed. Sensitivity analysis may be performed with data from all patients including data collected after discontinuing treatment up to week 16.

#### 10.4.4.2. Adverse Events

## **Definitions**

Treatment-emergent adverse events are defined as those that are not present at baseline or represent the exacerbation of a pre-existing condition during the on-treatment period.

## <u>Analysis</u>

All AEs reported in this study will be coded using the currently available version of the Medical Dictionary for Regulatory Activities (MedDRA®). Coding will be to lowest level terms. The verbatim text, the preferred term (PT), and the primary system organ class (SOC) will be listed. Post-treatment AEs and all AEs during the study will be summarized similarly as TEAEs.

Summaries of all TEAEs by treatment group will include:

- The number (n) and percentage (%) of patients with at least 1 TEAE by SOC and PT
- TEAEs by severity (according to the grading scale outlined in Section 9.5.1), presented by SOC and PT
- TEAEs by relationship to treatment (related, not related), presented by SOC and PT
- Treatment-emergent AESIs (defined with a PT or a prespecified grouping)

Deaths and other SAEs will be listed and summarized by treatment group.

Treatment-emergent adverse events leading to permanent treatment discontinuation will be listed and summarized by treatment group.

In addition, AESIs will be reported according to the adjudicated diagnosis. Imaging data related to AA including change from baseline in joint space width will be summarized.

## **10.4.4.3.** Other Safety

#### Vital Signs

Vital signs (temperature, pulse, blood pressure, and respiration rate) will be summarized by baseline and change from baseline to each scheduled assessment time with descriptive statistics.

#### Laboratory Tests

Laboratory test results will be summarized by baseline and change from baseline to each scheduled assessment time with descriptive statistics.

Number and percentage of patients with a PCSV at any post randomization time point will be summarized for each clinical laboratory test.

Shift tables based on baseline normal/abnormal and other tabular and graphical methods may be used to present the results for laboratory tests of interest.

Listings will be provided with flags indicating the out of laboratory range values.

#### 10.4.4.4. Treatment Exposure

Because of the half-life of the biologic being studied, the duration of fasinumab exposure during the study will be presented by treatment group and calculated as:

(Date of last administration of study drug - date of the first study drug administration after randomization) + 28

The number and percentage of patients randomized and exposed to double-blind study drug will be presented by specific time period for each treatment group.

## **10.4.4.5.** Treatment Compliance

Overall treatment compliance is defined as the actual dose of injection compared to the prescribed dose of treatment during the treatment period up to treatment discontinuation. It is calculated according to the following formula:

100\* Total actual injection dose taken/Prescribed injection dose.

The total number of actual doses of fasinumab will be summarized.

#### **10.4.5.** Analysis of Drug Concentration Data

Summaries of concentrations of functional fasinumab in serum will be presented descriptively by nominal time. Plots of individual concentration over time will be presented by actual day. Plots of mean or median concentrations of functional fasinumab will be presented by nominal day or week.

No formal statistical analysis will be performed.

## 10.4.6. Analysis of Anti-Drug Antibody Data

Immunogenicity will be characterized by the ADA response observed:

- Treatment-emergent ADA response defined as any post-dose positive ADA assay response when the baseline results are negative
- Treatment-boosted ADA response defined as any post-dose positive ADA assay response that is 9-fold over baseline titer levels when baseline is positive in the ADA assay
- Maximum ADA titer values
  - Low (titer < 1,000)
  - Moderate  $(1,000 \le \text{titer} \le 10,000)$
  - High (titer > 10,000)

Listings of ADA positivity and titers presented by patient, time point, and dose group will be provided. Incidence of treatment-emergent ADA response will be assessed as absolute occurrence (N) and percent of patients (%), grouped by study cohorts.

The influence of ADAs on drug concentrations will be evaluated. Assessment of impact of ADAs on safety and efficacy may be provided.

## 10.5. Interim Analysis

An interim analysis may be performed after 50% patients have completed the 16-week treatment period in order to assess peripheral nerve safety data for regulatory purposes.

## **10.6.** Additional Statistical Data Handling Conventions

The following analysis and data conventions will be followed:

General rules for handling missing data:

- Rules for handling missing data for efficacy assessments due to missing individual item data will follow each questionnaire's instrument manual.
- If the start date of an AE or concomitant medication is incomplete or missing, it will be assumed to have occurred on or after the intake of study medication, except if an incomplete date (eg, month and year) clearly indicates that the event started prior to treatment. If the partial date indicates the same month or year of the intake of study medication date, then the start date by the study medication intake date will be imputed; otherwise, the missing day or month by the first day or the first month will be imputed.
- No imputations for missing laboratory data, ECG data, vital sign data, or physical examination data will be made.

#### Visit windows:

• Assessments taken outside of protocol allowable windows will be displayed according to the CRF assessment recorded by the investigator.

#### Unscheduled assessments:

• Extra assessments (laboratory data or vital signs associated with nonprotocol clinical visits or obtained in the course of investigating or managing AEs) will be included in listings, but not summaries. If more than 1 laboratory value is available for a given visit, the first observation will be used in summaries and all observations will be presented in listings.

# 10.7. Statistical Considerations Surrounding the Premature Termination of a Study

If the study is terminated prematurely, only those parameters required for the development program and/or reporting to regulatory authorities will be summarized. Investigator and sponsor responsibilities surrounding the premature termination of a study are presented in Section 16.1.
#### 11. DATA MANAGEMENT AND ELECTRONIC SYSTEMS

## 11.1. Data Management

A data management plan specifying all relevant aspects of data processing for the study (including data validation, cleaning, correcting, releasing) will be maintained and stored at Regeneron.

A medical coding plan will specify the processes and the dictionary used for coding. All data coding (eg, AEs, baseline findings, medication, medical history, surgical history) will be done using internationally recognized and accepted dictionaries.

The eCRF data for this study will be collected with an electronic data capture (EDC) tool, Rave Medidata.

## 11.2. Electronic Systems

Electronic systems that may be used to process and/or collect data in this study will include the following:

- IWRS system randomization and study drug supply
- Rave Medidata EDC system clinical data capture
- Statistical Analysis System statistical review and analysis
- Argus pharmacovigilance and clinical safety software system for the collection and reporting of SAEs and AESIs
- Electronic Clinical Outcome Assessment systems collected patient-reported or patient clinical assessment results
- RAVE Medidata Imaging System electronic platform used to upload nerve conduction test wave forms for central reader review

## 12. STUDY MONITORING

# **12.1.** Monitoring of Study Sites

The study monitor and/or designee (eg, CRO monitor) will visit each site prior to enrollment of the first patient, and periodically during the study.

The investigator must allow study-related monitoring.

The study monitors will perform ongoing source data review to verify that data recorded in the CRF by authorized site personnel are accurate, complete, and verifiable from source documents, that the safety and rights of patients are being protected, and that the study is being conducted in accordance with the current approved protocol version and any other study agreements, ICH GCP, and all applicable regulatory requirements.

# **12.2.** Source Document Requirements

Investigators are required to prepare and maintain adequate and accurate patient records (source documents).

The investigator must keep all source documents on file with the CRF (throughout this protocol, CRF refers to either a paper CRF or an electronic CRF). Case report forms and source documents must be available at all times for inspection by authorized representatives of the sponsor and regulatory authorities.

## 12.3. Case Report Form Requirements

Study data obtained in the course of the clinical study will be recorded on electronic CRFs within the EDC system by trained site personnel. All required CRFs must be completed for each patient enrolled in the study. After review of the clinical data for each patient, the investigator must provide an electronic signature. A copy of each patient CRF casebook is to be retained by the investigator as part of the study record and must be available at all times for inspection by authorized representatives of the sponsor and regulatory authorities.

The investigator must ensure the accuracy, completeness, and timeliness of the data reported to the sponsor in the CRFs.

Corrections to the CRF will be entered in the CRF by the investigator or an authorized designee. All changes, including date and person performing corrections, will be available via the audit trail, which is part of the EDC system. For corrections made via data queries, a reason for any alteration must be provided.

#### 13. AUDITS AND INSPECTIONS

This study may be subject to a quality assurance audit or inspection by the sponsor or regulatory authorities. Should this occur, the investigator is responsible for:

- Informing the sponsor of a planned inspection by the authorities as soon as notification is received, and authorizing the sponsor's participation in the inspection
- Providing access to all necessary facilities, study data, and documents for the inspection or audit
- Communicating any information arising from inspection by the regulatory authorities to the sponsor immediately
- Taking all appropriate measures requested by the sponsor to resolve the problems found during the audit or inspection

Documents subject to audit or inspection include but are not limited to all source documents, CRFs, medical records, correspondence, ICFs, IRB or EC files, documentation of certification and quality control of supporting laboratories, and records relevant to the study maintained in any supporting pharmacy facilities. Conditions of study material storage are also subject to inspection. In addition, representatives of the sponsor may observe the conduct of any aspect of the clinical study or its supporting activities both within and outside of the investigator's institution.

In all instances, the confidentiality of the data must be respected.

## 14. ETHICAL AND REGULATORY CONSIDERATIONS

#### **14.1.** Good Clinical Practice Statement

It is the responsibility of both the sponsor and the investigator(s) to ensure that this clinical study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki, and that are consistent with the ICH guidelines for GCP and applicable regulatory requirements.

## 14.2. Informed Consent

The principles of informed consent are described in ICH guidelines for GCP.

The ICF used by the investigator must be reviewed and approved by the sponsor prior to submission to the appropriate IRB or EC. A copy of the IRB- or EC-approved ICF and documentation of approval must be provided to the sponsor before study drug will be shipped to the study site.

It is the responsibility of the investigator or designee (if acceptable by local regulations) to obtain written informed consent from each patient prior to his/her participation in the study and after the aims, methods, objectives, and potential hazards of the study have been explained to the patient in language that he/she can understand. The ICF should be signed and dated by the patient and by the investigator or authorized designee who reviewed the ICF with the patient.

- Patients who can write but cannot read will have the ICF read to them before signing and dating the ICF
- Patients who can understand but who can neither write nor read will have the ICF read to them in presence of an impartial witness, who will sign and date the ICF to confirm that informed consent was given

The original ICF must be retained by the investigator as part of the patient's study record, and a copy of the signed ICF must be given to the patient.

If new safety information results in significant changes in the risk/benefit assessment, the ICF must be reviewed and updated appropriately. All study patients must be informed of the new information and provide their written consent if they wish to continue in the study. The original signed revised ICF must be maintained in the patient's study record and a copy must be given to the patient.

# 14.3. Patient Confidentiality and Data Protection

The investigator must take all appropriate measures to ensure that the anonymity of each study patient will be maintained. Patients should be identified by their patient identification number, only, on CRFs or other documents submitted to the sponsor. Documents that will not be submitted to the sponsor (eg, signed ICF) must be kept in strict confidence.

The patient's identifiers and investigator's personal data, which may be included in the sponsor database, will be treated in compliance with all applicable laws and regulations. The sponsor shall take all appropriate measures to safeguard and prevent access to this data by any unauthorized third party.

#### 14.4. Institutional Review Board/Ethics Committee

An appropriately constituted IRB or EC, as described in ICH guidelines for GCP, must review and approve:

- The protocol, ICF, and any other materials to be provided to the patients (eg, advertising) before any patient may be enrolled in the study
- Any amendment or modification to the study protocol or ICF before implementation, unless the change is necessary to eliminate an immediate hazard to the patients, in which case the IRB or EC should be informed as soon as possible
- Ongoing studies on an annual basis or at intervals appropriate to the degree of risk

In addition, the IRB or EC should be informed of any event likely to affect the safety of patients or the continued conduct of the clinical study.

A copy of the IRB- or EC-approval letter with a current list of the IRB or EC members and their functions must be received by the sponsor prior to shipment of drug supplies to the investigator. The approval letter should include the study number and title, the documents reviewed, and the date of the review.

Records of the IRB or EC review and approval of all study documents (including approval of ongoing studies) must be kept on file by the investigator.

# 14.5. Clinical Study Data Transparency

Final study results will be published on a public clinical trial website according to applicable local guidelines and regulations. Treatment codes will be disseminated to each investigation site thereafter.

#### 15. PROTOCOL AMENDMENTS

The sponsor may not implement a change in the design of the protocol or ICF without an IRB- or EC-approved amendment. Regulatory approval will also be obtained where required by local regulations.

# 16. PREMATURE TERMINATION OF THE STUDY OR CLOSE-OUT OF A SITE

# **16.1.** Premature Termination of the Study

The sponsor has the right to terminate the study prematurely. Reasons may include efficacy, safety, or futility, among others. Should the sponsor decide to terminate the study, the investigator(s) will be notified in writing.

#### 16.2. Close-out of a Site

The sponsor and the investigator have the right to close-out a site prematurely.

#### Investigator's Decision

The investigator must notify the sponsor of a desire to close-out a site in writing, providing at least 30 days' notice. The final decision should be made through mutual agreement with the sponsor. Both parties will arrange the close-out procedures after review and consultation.

#### Sponsor's Decision

The sponsor will notify the investigator(s) of a decision to close-out a study site in writing. Reasons may include the following, among others:

- The investigator has received all items and information necessary to perform the study, but has not enrolled any patient within a reasonable period of time
- The investigator has violated any fundamental obligation in the study agreement, including but not limited to, breach of this protocol (and any applicable amendments), breach of the applicable laws and regulations, or breach of any applicable ICH guidelines
- The total number of patients required for the study are enrolled earlier than expected

In all cases, the appropriate IRB or EC and Health Authorities must be informed according to applicable regulatory requirements, and adequate consideration must be given to the protection of the patients' interests.

#### 17. STUDY DOCUMENTATION

# 17.1. Certification of Accuracy of Data

A declaration assuring the accuracy and content of the data recorded on the eCRF must be signed electronically by the investigator. This signed declaration accompanies each set of patient final eCRF that will be provided to the sponsor.

## 17.2. Retention of Records

The investigator must retain all essential study documents, including ICFs, source documents, investigator copies of CRFs, and drug accountability records for at least 15 years following the completion or discontinuation of the study, or longer, if a longer period is required by relevant regulatory authorities. The investigator must obtain written approval from the sponsor before discarding or destroying any essential study documents during the retention period following study completion or discontinuation. Records must be destroyed in a manner that ensures confidentiality.

If the investigator's personal situation is such that archiving can no longer be ensured, the investigator must inform the sponsor (written notification) and the relevant records will be transferred to a mutually agreed-upon destination.

# 18. DATA QUALITY ASSURANCE

In accordance with ICH E6, the sponsor is responsible for quality assurance to ensure that the study is conducted and the data generated, recorded, and reported in compliance with the protocol,

GCP, and any applicable regulatory requirement(s). The planned quality assurance and quality control procedures for the study are summarized.

## Data Management

The sponsor is responsible for the data management of this study including quality checking of the data (Section 11.1).

## Study Monitoring

The investigator must allow study-related monitoring, IRB/EC review, audits, and inspections from relevant health regulatory authorities, and provide direct access to source data documents (Section 12.1, Section 12.2, and Section 13).

The study monitors will perform ongoing source data review to verify that data recorded in the CRF by authorized site personnel are accurate, complete, and verifiable from source documents, that the safety and rights of patients are being protected, and that the study is being conducted in accordance with the current approved protocol version and any other study agreements, ICH GCP, and all applicable regulatory requirements (Section 12.1).

All patient data collected during the study will be recorded on paper or electronic CRF unless the data are transmitted to the sponsor or designee electronically (eg, laboratory data). The investigator is responsible for affirming that data entries in the CRF are accurate and correct by electronically signing a declaration that accompanies each set of patient final CRF (Section 12.3, Section 17.1).

#### **Study Documentation**

The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF (Section 12.2).

The investigator will retain all records and documents, including signed ICFs, pertaining to the conduct of this study for at least 15 years after study completion, unless local regulations or institutional policies require a longer retention period. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor (Section 17.2).

#### 19. CONFIDENTIALITY

Confidentiality of information is provided as a separate agreement.

#### 20. FINANCING AND INSURANCE

Financing and insurance information is provided as a separate agreement.

#### 21. PUBLICATION POLICY

The publication policy is provided as a separate agreement.

#### 22. REFERENCES

Aloe, L., M.A. Tuveri, U. Carcassi, and R. Levi-Montalcini. Nerve growth factor in the synovial fluid of patients with chronic arthritis. Arthritis Rheum. 1992. 35:351-355.

Altman, R., G. Alarcon, D. Appelrouth, D. Bloch, D. Borenstein, K. Brandt, C. Brown, T.D. Cooke, W. Daniel, D. Feldman, and et al. The American College of Rheumatology criteria for the classification and reporting of osteoarthritis of the hip. Arthritis Rheum. 1991. 34:505-514.

Altman, R., E. Asch, D. Bloch, G. Bole, D. Borenstein, K. Brandt, W. Christy, T.D. Cooke, R. Greenwald, M. Hochberg, and et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986. 29:1039-1049. Available at:

http://www.rheumatology.org/Portals/1030/Files/Complete%1020Article\_Osteoarthritis%1020of%1020the%1020Knee%1020-%201986.pdf.

Arezzo JC, Rosenstock J, LaMoreaux L, Pauer L. Efficacy and safety of pregabalin 600 mg/d for treating painful diabetic peripheral neuropathy: A double-blind placebo-controlled trial. BMC Neurology 2008. 8:33

Bingham, C.O., 3rd, A.I. Sebba, B.R. Rubin, G.E. Ruoff, J. Kremer, S. Bird, S.S. Smugar, B.J. Fitzgerald, K. O'Brien, and A.M. Tershakovec. Efficacy and safety of etoricoxib 30 mg and celecoxib 200 mg in the treatment of osteoarthritis in two identically designed, randomized, placebo-controlled, non-inferiority studies. Rheumatology (Oxford). 2007. 46:496-507.

Bjordal, J.M., A.E. Ljunggren, A. Klovning, and L. Slordal. Non-steroidal anti-inflammatory drugs, including cyclo-oxygenase-2 inhibitors, in osteoarthritic knee pain: meta-analysis of randomised placebo controlled trials. BMJ. 2004. 329:1317.

Brown, M.T., F.T. Murphy, D.M. Radin, I. Davignon, M.D. Smith, and C.R. West. Tanezumab reduces osteoarthritic knee pain: results of a randomized, double-blind, placebo-controlled phase III trial. J Pain. 2012. 13:790-798.

Chao, M.V., R. Rajagopal, and F.S. Lee. Neurotrophin signaling in health and disease. Clinical Science. 2006. 110:167-173.

Crowley, C., S.D. Spencer, M.C. Nishimura, K.S. Chen, S. Pitts-Meek, M.P. Armanini, L.H. Ling, S.B. McMahon, D.L. Shelton, A.D. Levinson, and et al. Mice lacking nerve growth factor display perinatal loss of sensory and sympathetic neurons yet develop basal forebrain cholinergic neurons. Cell. 1994. 76:1001-1011.

Dibonaventura, M., S. Gupta, M. McDonald, and A. Sadosky. Evaluating the health and economic impact of osteoarthritis pain in the workforce: results from the National Health and Wellness Survey. BMC Musculoskelet Disord. 2011. 12:83.

Dolgin, M., Editor. 1994. Nomenclature and Criteria for Diagnosis of Diseases of the Heart and Great Vessels. In The Criteria Committee of the New York Heart Association, 9th Edition. Little, Brown, and Co., Boston, MA. 253-256.

Einarsdottir, E., A. Carlsson, J. Minde, G. Toolanen, O. Svensson, G. Solders, G. Holmgren, D. Holmberg, and M. Holmberg. A mutation in the nerve growth factor beta gene (NGFB) causes loss of pain perception. Hum Mol Genet. 2004. 13:799-805.

Halliday, D.A., C. Zettler, R.A. Rush, R. Scicchitano, and J.D. McNeil. Elevated nerve growth factor levels in the synovial fluid of patients with inflammatory joint disease. Neurochem Res. 1998. 23:919-922.

Harris, W.H. Traumatic arthritis of the hip after dislocation and acetabular fractures: treatment by mold arthroplasty. An end-result study using a new method of result evaluation. J Bone Joint Surg Am. 1969. 51:737-755.

Hefti, F., M. Mokhtarani, M. Gray, C. Zhao, and C. Chan. RN624 (Anti-NGF) reduces pain and improves function in subjects with moderate to severe pain form osteoarthritis of the knee. The Journal of Pain. 2006. 7:S46.

Indo, Y., M. Tsuruta, Y. Hayashida, M.A. Karim, K. Ohta, T. Kawano, H. Mitsubuchi, H. Tonoki, Y. Awaya, and I. Matsuda. Mutations in the TRKA/NGF receptor gene in patients with congenital insensitivity to pain with anhidrosis. Nat Genet. 1996. 13:485-488.

Insall, J.N., L.D. Dorr, R.D. Scott, and W.N. Scott. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989.13-14.

Katz, N., D.G. Borenstein, C. Birbara, C. Bramson, M.A. Nemeth, M.D. Smith, and M.T. Brown. Efficacy and safety of tanezumab in the treatment of chronic low back pain. Pain. 2011. 152:2248-2258.

Kivitz, AJ, J.S. Gimbel, C. Bramson, M.A. Nemeth, D.S. Keller, M.T. Brown, C.R. West, and K.M. Verburg. Efficacy and safety of tanezumab versus naproxen in the treatment of chronic low back pain. Pain. 2013. 154:1009-1021.

Lanas, A. Gastrointestinal bleeding associated with low-dose aspirin use: relevance and management in clinical practice. Expert Opin Drug Saf. 2011. 10:45-54.

Lane, N.E., T.J. Schnitzer, C.A. Birbara, M. Mokhtarani, D.L. Shelton, M.D. Smith, and M.T. Brown. Tanezumab for the treatment of pain from osteoarthritis of the knee. N Engl J Med. 2010. 363:1521-1531.

Lewin, G.R., A. Rueff, and L.M. Mendell. Peripheral and central mechanisms of NGF-induced hyperalgesia. Eur J Neurosci. 1994. 6:1903-1912.

Liu S, Blanchard S, Bigou S, Vitry S, Bohl D, Heard JM. Neurotrophin 3 improves delayed reconstruction of sensory pathways after cervical dorsal root injury. Neurosurgery. 2011 Feb;68(2):450-61

Lowe, E.M., P. Anand, G. Terenghi, R.E. Williams-Chestnut, D.V. Sinicropi, and J.L. Osborne. Increased nerve growth factor levels in the urinary bladder of women with idiopathic sensory urgency and interstitial cystitis. Br J Urol. 1997. 79:572-577.

Makarowski, W., W.W. Zhao, T. Bevirt, and D.P. Recker. Efficacy and safety of the COX-2 specific inhibitor valdecoxib in the management of osteoarthritis of the hip: a randomized, double-blind, placebo-controlled comparison with naproxen. Osteoarthritis Cartilage. 2002. 10:290-296.

Mallik A, Weir AI. Nerve conduction studies: Essentials and pitfalls in practice. J Neurol Neurosurg Psychiatry. 2005. 76(Suppl II): ii23-ii31.

McArthur, JC, Yiannoutsos C, Simpson D, Adornato BT, Singer EJ, Hollander H, et al. A phase II trial of nerve growth factor for sensory neuropathy associated with HIV infection. AIDS Clinical Trials Group Team 291. Neurology. 2000. 54:1080-1088.

Miller LJ, Fischer KA, Goralnick SJ, MLitt M, Burleson JA, PAlbertsen P, et al. Nerve growth factor and chronic prostatitis/chronic pelvic pain syndrome. Urology. 2002. 59:603-608.

Parkman HP, Rao SS, Reynolds JC, Schiller LR, Wald A, Miner PB et al. Neurotrophin-3 improves functional constipation. Am J Gastroenterol. 2003 Jun;98(6):1338-47.

Pezet S, McMahon SB. Neurotrophins: mediators and modulators of pain. Annu Rev Neurosci. 2006. 29:507-538.

Ramer MS, Bisby MA. Adrenergic innervation of rat sensory ganglia following proximal or distal painful sciatic neuropathy: distinct mechanisms revealed by anti-NGF treatment. Eur J Neurosci. 1999. 11:837-846.

Salmon JH, Rat AC, Sellam J, Michel M, Eschard JP, Guillemin F, et al. Economic impact of lower-limb osteoarthritis worldwide: a systematic review of cost-of-illness studies. Osteoarthritis Cartilage. 2016. 24:1500-1508.

Sarchielli P, Alberti A, Floridi A, Gallai V. Levels of nerve growth factor in cerebrospinal fluid of chronic daily headache patients. Neurology. 2001. 57:132-134.

Sarzi-Puttini P, Cimmino MA, Scarpa R, RCaporali R, Parazzini F, Zaninelli A, et al. Osteoarthritis: an overview of the disease and its treatment strategies. Semin Arthritis Rheum. 2005. 35:1-10.

Silverstein FE, Faich G, Goldstein JL, Simon LS, Pincus T, Whelton A, et al. Gastrointestinal toxicity with celecoxib vs nonsteroidal anti-inflammatory drugs for osteoarthritis and rheumatoid arthritis: the CLASS study: A randomized controlled trial. Celecoxib Long-term Arthritis Safety Study. JAMA. 2000. 284:1247-1255.

Smeyne RJ, Klein R, Schnapp A, Long LK, Bryant S, Lewin A, et al. Severe sensory and sympathetic neuropathies in mice carrying a disrupted Trk/NGF receptor gene. Nature. 1994. 368:246-249.

Trelle S, Reichenbach S, Wandel S, Hildebrand P, Tschannen B, Villiger PM, et al. Cardiovascular safety of non-steroidal anti-inflammatory drugs: network meta-analysis. BMJ. 2011. 342:c7086.

#### 23. INVESTIGATOR'S AGREEMENT

I have read the attached protocol, entitled "A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Effects of Fasinumab on Peripheral Nerve Function in Patients with Pain due to Osteoarthritis of the Knee or Hip," dated as noted in the appended signature page, and agree to abide by all provisions set forth therein.

I agree to comply with the current International Council for Harmonisation Guideline for Good Clinical Practice and the laws, rules, regulations, and guidelines of the community, country, state, or locality relating to the conduct of the clinical study.

I also agree that persons debarred from conducting or working on clinical studies by any court or regulatory agency will not be allowed to conduct or work on studies for the sponsor or a partnership in which the sponsor is involved. I will immediately disclose it in writing to the sponsor if any person who is involved in the study is debarred, or if any proceeding for debarment is pending, or, to the best of my knowledge, threatened.

This document contains confidential information of the sponsor, which must not be disclosed to anyone other than the recipient study staff and members of the Institutional Review Board or Ethics Committee. I agree to ensure that this information will not be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of the sponsor.

| (Signature of Investigator) | (Date) |
|-----------------------------|--------|
| (Printed Name) | |

#### SIGNATURE OF SPONSOR'S RESPONSIBLE OFFICERS

(Medical/Study Director, Regulatory Representative, Clinical Study Team Lead, and Biostatistician)

To the best of my knowledge, this report accurately describes the conduct of the study.

Study Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to

Evaluate the Effects of Fasinumab on Peripheral Nerve Function in Patients

with Pain Due to Osteoarthritis of the Hip or Knee

Protocol Number: R475-OA-1758

Protocol Version: R475-OA-1758 Amendment 2

See appended electronic signature page

Sponsor's Responsible Medical/Study Director

See appended electronic signature page

Sponsor's Responsible Regulatory Liaison

See appended electronic signature page

Sponsor's Responsible Clinical Study Team Lead

See appended electronic signature page

Sponsor's Responsible Biostatistician

Signature Page for VV-RIM-00063020 v2.0



Signature Page for VV-RIM-00063020 v2.0 Approved